CLINICAL TRIAL: NCT01362244
Title: A Randomised, Double-Blind, Placebo Controlled, Multi-Center Study To Investigate The Use Of Mepolizumab (Sb-240563) In Reducing The Need For Surgery In Subjects With Severe Bilateral Nasal Polyposis
Brief Title: Mepolizumab in Nasal Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111782; 2008-003772-21 (EudraCT Number)
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Nasal Polyps
Keywords: Quality of Life; Intranasal Steroids; Severe Nasal Polyposis; Polyp Relapse; Endoscopic Polyp Score; Surgery
MeSH Terms: conditions — Nasal Polyps | interventions — mepolizumab; Jogging; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Periods 1-8 (Experimental): Part A comprises eight outpatient visits (Visits 1 - 8). For six of these visits, subjects will receive a dose of either 750 mg mepolizumab or placebo. Dosing occurs in four week intervals. Assessment for entry into Part B will take place at the last visit in Part A (Visit 8). Subjects not eligible for Part B will have study exit procedures performed and be discontinued.
  Interventions: Drug: Mepolizumab; Drug: Placebo
- Run In period (Other): 10-14 day run in period to assess the patients suitability for entry into Part A of the trial.
  Interventions: Drug: Run In Medication
- Treatment periods 9-13 (No Intervention): Subjects eligible for Part B will attend the clinic for up to 5 more outpatient visits (Visits 9 - 13) for assessments. Visits occur every four weeks. There is no dosing in Part B. At the point when each subject meets Study Exit criteria, study exit procedures will be performed and the subject will exit the study.

INTERVENTIONS:
Drug: Mepolizumab — 750 mg of mepolizumab by IV infusion
  Arms: Treatment Periods 1-8
Drug: Placebo — Placebo by IV infusion
  Arms: Treatment Periods 1-8
Drug: Run In Medication — subjects will undergo a run-in period of 10 - 14 days on a low dose of Intranasal Steroids (INS).
  Arms: Run In period

SUMMARY:
A two-part, randomised, double-blind, placebo controlled, multi-centre study to investigate the use of mepolizumab (SB-240563) in reducing the need for surgery in subjects with severe bilateral nasal polyposis.

DETAILED DESCRIPTION:
Nasal polyposis has long been known as chronic inflammatory disease of the nasal mucosa. This disease is characterized by the presence of polyps in the upper nasal cavity, originating from within the ostiomeatal complex. The presence of polyps can cause long-term symptoms such as prominent nasal obstruction, post-nasal drip, loss of smell, and discharge. These symptoms can impact greatly upon a patient's quality of life.The etiology of nasal polyposis is currently unknown.

The aim of this present study is to investigate the use of mepolizumab in reducing the potential need for surgery in subjects with severe bilateral nasal polyposis. The study is split into two parts: Part A is the treatment phase and focuses on the reduction of the need for surgery by exploring the efficacy of six doses of mepolizumab (one dose every four weeks) on nasal polyposis. This dosing regime will build upon the previous PoC study by exploring the potential for increased clinical efficacy as assessed by the potential need for surgery, and also and increased duration of action as assessed by time to relapse. Part B is the follow-up phase and will assess post-treatment nasal polyposis dynamics with a focus on time to relapse. All subjects participating in this study will undergo a run-in period on a low dose of intranasal steroids (INS) prior to first dosing. INS will be continued throughout the study up until study exit. This is to reflect the real life circumstances in which mepolizumab is intended to be used as a therapy. The overall aim of the study design is to further assess the impact in the potential need for surgery and explore an appropriate mepolizumab therapeutic regimen strategy for the treatment of nasal polyposis.

In this study, the assessment of nasal polyposis will be performed by means of combining endoscopic polyp score with subject reported symptoms. This approach reflects real-life clinical assessment of nasal polyposis. Also, this study incorporates condition specific and general medical questionnaires in order to obtain a better understanding of the impact of severe nasal polyposis of the subject's quality of life (QOL). This is in line with increasing focus in the medical field on the effects of medical conditions and treatments on the quality of life of patients (Fokkens et al 2007).

ELIGIBILITY:
Inclusion:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Subjects have a diagnosis of severe bilateral nasal polyposis at the screening visit and Visit 1 (i.e. at end of run-in period) which meets the definition of the situation indicative of the need for surgery as described in Decision Table 1 in Appendix 3.
2. Subjects must have had at least one previous surgery for the removal of nasal polyps.
3. Subjects must have an history of refractory response to steroid therapy as shown by being deemed potentially eligible for surgery despite having been on a regular/continuous course of nasal corticosteroids for the treatment of nasal polyposis for at least 3 months and/or have received a short course of oral steroids in the past for nasal polyp treatment.
4. Male or female between 18 and 70 years of age, inclusive at time of signing informed consent.
5. BMI within the range 19.0 to 31.0 kg/m2 (inclusive).
6. Subjects must be free of any clinically significant disease that would interfere with the study schedule or procedures or compromise his/her safety.
7. Subjects with concurrent asthma must be maintained on no more than 10mg/day of Prednisolone or the equivalent.
8. Female subjects of childbearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from 1 month prior to first dose of study medication until four months after last dose of study medication.

   Females of non -childbearing potential are defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study (from 1 month prior to first dose of study medication until four months after last dose of study medication). Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2- 4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
9. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until four months after last dose of study medication.
10. Subjects are capable of giving written informed consent, which includes agreeing to be compliant with the study requirements and restrictions listed in the consent form.
11. Subjects are willing and available to complete the study and all measurements.
12. Subjects are capable of reading, comprehending, and writing the local language at a sufficient level to complete study related materials.

Exclusion:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. As a result of medical interview, physical examination, or screening investigation the physician responsible considers the subject unfit for the study.
2. Subjects requiring oral corticosteroids at a dose greater than 10mg Prednisolone or equivalent during the study will be terminated from the study.
3. Subjects who have had an asthma exacerbation requiring admission to hospital within 4 weeks of Screening.
4. Subjects who have received immunotherapy within the previous 12 months.
5. Subjects with a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
6. Subjects with a known medical history of Hepatitis B, Hepatitis C, or HIV infection.
7. Subjects with a history or suspicion of drug abuse or alcohol abuse within the last 6 months.
8. Subjects who are currently receiving, or have received within 3 months prior to first mepolizumab dose, chemotherapy, radiotherapy or investigational medications/therapies.
9. Subjects with one or more of the following abnormal laboratory values:

   * Serum creatinine ≥ 3 times institutional ULN
   * AST or/ALT ≥ 5 times institutional ULN
   * Platelet count < 50,000/μL
10. Subjects with a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. Aspirin-sensitive subjects are acceptable.
11. Subjects with a history of allergic reaction to anti-IL-5 or other antibody therapy.
12. Pregnant females as determined by positive serum pregnancy test at screening or positive urine pregnancy test prior to each dosing occasion.
13. Breastfeeding/Lactating females.
14. Subjects who currently smoke or have smoked in the last 6 months.
15. Subjects who are unwilling or unable to follow the procedures outlined in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-05-12 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2014-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Ghent, Belgium
- GSK Investigational Site, Amsterdam, Netherlands
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bachert C, Sousa AR, Lund VJ, Scadding GK, Gevaert P, Nasser S, Durham SR, Cornet ME, Kariyawasam HH, Gilbert J, Austin D, Maxwell AC, Marshall RP, Fokkens WJ. Reduced need for surgery in severe nasal polyposis with mepolizumab: Randomized trial. J Allergy Clin Immunol. 2017 Oct;140(4):1024-1031.e14. doi: 10.1016/j.jaci.2017.05.044. Epub 2017 Jul 4. PMID 28687232
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111782 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the end of a 10- to 14-day Run-in Period, participants (par.) were assessed for entry into the Treatment Period, comprised of 8 outpatient visits. For 6 of these visits, participants received a 4-weekly dose of either 750 milligrams (mg) mepolizumab or placebo. Four of the par. withdrew prior to 1st dose and are not included in the par. flow.
Groups:
- Mepolizumab 750 mg: Participants received up to a total of six doses (one every 4 weeks) of mepolizumab 750 milligrams (mg) by intravenous infusion.
- Placebo: Participants received up to a total of six doses (one every 4 weeks) of matching placebo by intravenous infusion.
Period: Overall Study
Arm/Group | Mepolizumab 750 mg | Placebo
Started | 54 | 51
Completed | 22 | 19
Not Completed | 32 | 32
Not completed — Adverse Event | 3 | 5
Not completed — Lack of Efficacy | 5 | 11
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Did not Meet Continuation Criteria | 17 | 11
Not completed — Protocol Defined Stopping Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepolizumab 750 mg | Placebo | Total
Number analyzed (Participants) | 54 | 51 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.6 (10.73) | 49.7 (10.38) | 50.2 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 41 | 34 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Central/South Asian Heritage (Htg) | 2 | 0 | 2
  Japanese/East Asian Heritage/ South East Asian Htg | 0 | 1 | 1
  White | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduced Need for Surgery at Week 25
Description: Assessment of the nasal polyposis condition was performed after six months of dosing to determine the situation indicative of a reduction in the need for surgery. The components used to determine the need for surgery were endoscopic polyp (ENP) scores and a severity of condition as measured by a visual analogue scale (VAS). Surgery was still deemed required for a participant with an ENP score of >=3, or an ENP score of 2 and a VAS symptom score of >7. The number of participants with reduced need for polyp surgery are presented as missing data set to non-responders (NR) and missing data last observation carry forward (LOCF). LOCF is defined as missing responses at Week 25 imputed with the last non-missing post-dose observation for that participant.
Time Frame: Week 25
Population: Per Protocol Population: all randomized participants who received at least one dose of study treatment and who complied with the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 49 | 51
Participants
  NR, Responders | 16 | 5
  NR, Non-Responders | 33 | 46
  LOCF, Responders | 17 | 8
  LOCF, Non- Responders | 32 | 43
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Statistical data is presented for NR; Test type: Superiority or Other; p = 0.003, Fisher Exact
Statistical Analysis 2: Comparison: Mepolizumab 750 mg vs Placebo; Statistical data is presented for LOCF; Test type: Superiority or Other; p = 0.016, Fisher Exact

2. Secondary Outcome: Number of Participants With Endoscopic Nasal Polyp (ENP) Score Dynamics at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Each nostril was assessed for polyps and graded at Weeks 1, 2, 5, 9, 13, 17, 21, and 25. The right and left nostrils were scored from 0 to 4, where, 0 = No polyps; 1 = Small polyps in the middle meatus not reaching below the inferior border of the middle concha; 2 = Polyps reaching below the lower border of the middle turbinate; 3 = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle concha; and 4 = Large polyps causing complete obstruction/congestion of the inferior meatus. The ENP score was recorded for both the right and the left nostril. The higher of the two scores was derived and used for the analysis. The ENP score ranges from 0 to 4, with a higher score indicating a larger polyp.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Population: PP Population. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 49 | 51
Participants
  Week 1, ENP score 0, n=49, 51 | 0 | 0
  Week 1, ENP score 1, n=49, 51 | 0 | 0
  Week 1, ENP score 2, n=49, 51 | 0 | 0
  Week 1, ENP score >=3, n=49, 51 | 49 | 51
  Week 2, ENP score 0, n=48, 51: number analyzed (Participants) | 48 | 51
  Week 2, ENP score 0, n=48, 51 | 0 | 0
  Week 2, ENP score 1, n=48, 51: number analyzed (Participants) | 48 | 51
  Week 2, ENP score 1, n=48, 51 | 0 | 0
  Week 2, ENP score 2, n=48, 51: number analyzed (Participants) | 48 | 51
  Week 2, ENP score 2, n=48, 51 | 1 | 0
  Week 2, ENP score >=3, n=48, 51: number analyzed (Participants) | 48 | 51
  Week 2, ENP score >=3, n=48, 51 | 47 | 51
  Week 5, ENP score 0, n=49, 48: number analyzed (Participants) | 49 | 48
  Week 5, ENP score 0, n=49, 48 | 0 | 0
  Week 5, ENP score 1, n=49, 48: number analyzed (Participants) | 49 | 48
  Week 5, ENP score 1, n=49, 48 | 0 | 0
  Week 5, ENP score 2, n=49, 48: number analyzed (Participants) | 49 | 48
  Week 5, ENP score 2, n=49, 48 | 8 | 6
  Week 5, ENP score >=3, n=49, 48: number analyzed (Participants) | 49 | 48
  Week 5, ENP score >=3, n=49, 48 | 41 | 42
  Week 9, ENP score 0, n=49, 45: number analyzed (Participants) | 49 | 45
  Week 9, ENP score 0, n=49, 45 | 0 | 0
  Week 9, ENP score 1, n=49, 45: number analyzed (Participants) | 49 | 45
  Week 9, ENP score 1, n=49, 45 | 5 | 0
  Week 9, ENP score 2, n=49, 45: number analyzed (Participants) | 49 | 45
  Week 9, ENP score 2, n=49, 45 | 8 | 5
  Week 9, ENP score >=3, n=49, 45: number analyzed (Participants) | 49 | 45
  Week 9, ENP score >=3, n=49, 45 | 36 | 40
  Week 13, ENP score 0, n=44, 37: number analyzed (Participants) | 44 | 37
  Week 13, ENP score 0, n=44, 37 | 3 | 0
  Week 13, ENP score 1, n=44, 37: number analyzed (Participants) | 44 | 37
  Week 13, ENP score 1, n=44, 37 | 5 | 0
  Week 13, ENP score 2, n=44, 37: number analyzed (Participants) | 44 | 37
  Week 13, ENP score 2, n=44, 37 | 5 | 2
  Week 13, ENP score >=3, n=44, 37: number analyzed (Participants) | 44 | 37
  Week 13, ENP score >=3, n=44, 37 | 31 | 35
  Week 17, ENP score 0, n=43, 34: number analyzed (Participants) | 43 | 34
  Week 17, ENP score 0, n=43, 34 | 3 | 1
  Week 17, ENP score 1, n=43, 34: number analyzed (Participants) | 43 | 34
  Week 17, ENP score 1, n=43, 34 | 4 | 1
  Week 17, ENP score 2, n=43, 34: number analyzed (Participants) | 43 | 34
  Week 17, ENP score 2, n=43, 34 | 7 | 6
  Week 17, ENP score >=3, n=43, 34: number analyzed (Participants) | 43 | 34
  Week 17, ENP score >=3, n=43, 34 | 29 | 26
  Week 21, ENP score 0, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, ENP score 0, n=42, 34 | 4 | 1
  Week 21, ENP score 1, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, ENP score 1, n=42, 34 | 6 | 2
  Week 21, ENP score 2, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, ENP score 2, n=42, 34 | 5 | 4
  Week 21, ENP score >=3, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, ENP score >=3, n=42, 34 | 27 | 27
  Week 25, ENP score 0, n=42, 31: number analyzed (Participants) | 42 | 31
  Week 25, ENP score 0, n=42, 31 | 3 | 1
  Week 25, ENP score 1, n=42, 31: number analyzed (Participants) | 42 | 31
  Week 25, ENP score 1, n=42, 31 | 7 | 2
  Week 25, ENP score 2, n=42, 31: number analyzed (Participants) | 42 | 31
  Week 25, ENP score 2, n=42, 31 | 7 | 4
  Week 25, ENP score >=3, n=42, 31: number analyzed (Participants) | 42 | 31
  Week 25, ENP score >=3, n=42, 31 | 25 | 24
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.710, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.15 to 3.64] — Week 1
Statistical Analysis 2: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.674, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.29 to 6.87] — Week 2
Statistical Analysis 3: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.942, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.20 to 4.49] — Week 5
Statistical Analysis 4: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.091, Regression, Logistic; Odds Ratio (OR) = 3.90, 95% CI 2-sided [0.80 to 18.96] — Week 9
Statistical Analysis 5: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 11.66, 95% CI 2-sided [2.18 to 62.33] — Week 13
Statistical Analysis 6: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.224, Regression, Logistic; Odds Ratio (OR) = 2.74, 95% CI 2-sided [0.54 to 13.90] — Week 17
Statistical Analysis 7: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 5.85, 95% CI 2-sided [1.11 to 30.69] — Week 21
Statistical Analysis 8: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.051, Regression, Logistic; Odds Ratio (OR) = 5.22, 95% CI 2-sided [0.99 to 27.44] — Week 25

3. Secondary Outcome: Number of Participants Who Required Polyp Surgery at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Assessment of the nasal polyposis condition was performed after 6 months of dosing to determine the situation indicative of a reduction in the need for surgery. The components used to determine the need for surgery were endoscopic polyp scores and a severity of condition as measured by a VAS. Surgery was required for participants with ENP scores of >=3, or ENP scores of 2 and a VAS symptom score of >7.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Population: PP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 49 | 51
Participants
  Week 1 | 49 | 51
  Week 2 | 48 | 51
  Week 5 | 44 | 49
  Week 9 | 39 | 48
  Week 13 | 38 | 50
  Week 17 | 37 | 46
  Week 21 | 35 | 46
  Week 25 | 33 | 46

4. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Weeks 2, 5, 9, 13, 17, 21, and 25
Description: SBP and DBP were measured at Baseline (Week 1) and at Weeks 2, 5, 9, 13, 17, 21, and 25. Baseline is defined as the Week 1 pre-dose assessment. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and Weeks 2, 5, 9, 13, 17, 21, and 25
Population: Safety Population: participants who received >=1 dose of study treatment (based on actual treatment received). One participant randomized to mepolizumab took placebo in error. Thus, "N" for the placebo arm of the SP is greater than for the ITT Population. Participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
millimeters of mercury (mmHg)
  SBP, Week 2, n=53, 52 | -2.0 (14.14) | 4.6 (13.33)
  SBP, Week 5, n=53, 49: number analyzed (Participants) | 53 | 49
  SBP, Week 5, n=53, 49 | -1.2 (11.74) | 0.5 (10.50)
  SBP, Week 9, n=51, 46: number analyzed (Participants) | 51 | 46
  SBP, Week 9, n=51, 46 | -0.9 (15.01) | 1.0 (12.84)
  SBP, Week 13, n=45, 40: number analyzed (Participants) | 45 | 40
  SBP, Week 13, n=45, 40 | -2.9 (12.17) | 0.9 (11.97)
  SBP, Week 17, n=45, 36: number analyzed (Participants) | 45 | 36
  SBP, Week 17, n=45, 36 | -1.9 (13.15) | 0.3 (11.72)
  SBP, Week 21, n=42, 34: number analyzed (Participants) | 42 | 34
  SBP, Week 21, n=42, 34 | -2.0 (14.55) | -1.7 (12.14)
  SBP, Week 25, n=42, 32: number analyzed (Participants) | 42 | 32
  SBP, Week 25, n=42, 32 | -2.4 (15.47) | -1.8 (15.39)
  DBP, Week 2, n=53, 52 | -1.3 (7.97) | -0.9 (10.44)
  DBP, Week 5, n=53, 49: number analyzed (Participants) | 53 | 49
  DBP, Week 5, n=53, 49 | 0.0 (8.56) | -0.1 (7.98)
  DBP, Week 9, n=51, 46: number analyzed (Participants) | 51 | 46
  DBP, Week 9, n=51, 46 | -1.8 (12.05) | 0.0 (7.29)
  DBP, Week 13, n=45, 40: number analyzed (Participants) | 45 | 40
  DBP, Week 13, n=45, 40 | -0.6 (9.99) | -0.5 (9.56)
  DBP, Week 17, n=45, 36: number analyzed (Participants) | 45 | 36
  DBP, Week 17, n=45, 36 | -2.2 (8.90) | -0.4 (9.43)
  DBP, Week 21, n=42, 34: number analyzed (Participants) | 42 | 34
  DBP, Week 21, n=42, 34 | -0.3 (7.95) | -1.5 (9.32)
  DBP, Week 25, n=42, 32: number analyzed (Participants) | 42 | 32
  DBP, Week 25, n=42, 32 | -1.5 (10.27) | -2.2 (9.58)

5. Secondary Outcome: Mean Change From Baseline in Pulse Rate at Weeks 2, 5, 9, 13, 17, 21, and 25
Description: Pulse rate was measured at Baseline (Week 1) and at Weeks 2, 5, 9, 13, 17, 21, and 25. Baseline is defined as the Week 1 pre-dose assessment. Change from Baseline is defined as the difference between the post-dose post-Baseline visit value and the Baseline value.
Time Frame: Baseline and Weeks 2, 5, 9, 13, 17, 21, and 25
Population: Safety Population. One participant randomized to mepolizumab took placebo in error. Thus, "N" for the placebo arm of the SP is greater than for the ITT Population. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
beats per minute
  Week 2, n=53, 52 | 0.2 (8.88) | 0.0 (7.86)
  Week 5, n=53, 50: number analyzed (Participants) | 53 | 50
  Week 5, n=53, 50 | -1.1 (9.09) | -1.0 (7.91)
  Week 9, n=51, 46: number analyzed (Participants) | 51 | 46
  Week 9, n=51, 46 | -1.7 (8.40) | -0.8 (7.50)
  Week 13, n=45, 40: number analyzed (Participants) | 45 | 40
  Week 13, n=45, 40 | -0.4 (11.05) | -2.4 (9.42)
  Week 17, n=45, 36: number analyzed (Participants) | 45 | 36
  Week 17, n=45, 36 | -0.4 (9.71) | -0.6 (9.35)
  Week 21, n=41, 34: number analyzed (Participants) | 41 | 34
  Week 21, n=41, 34 | -2.0 (9.56) | -1.2 (8.70)
  Week 25, n=41, 32: number analyzed (Participants) | 41 | 32
  Week 25, n=41, 32 | -0.4 (9.29) | 0.0 (8.29)

6. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: A single safety 12-lead ECG was performed using a standard 12-lead ECG machine at Weeks 1, 2, 5, 9, 13, 17, 21, and 25. Any abnormal clinically significant (CS) and not clinically significant (NCS) findings were identified. ECG abnormaility with respect to CS and NCS findings were judged by the investigator or appropriately qualified designee. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Week 1, NCS, n=53, 52 | 8 | 8
  Week 1, CS, n=53, 52 | 0 | 0
  Week 2, NCS, n=52, 52: number analyzed (Participants) | 52 | 52
  Week 2, NCS, n=52, 52 | 7 | 9
  Week 2, CS, n=52, 52: number analyzed (Participants) | 52 | 52
  Week 2, CS, n=52, 52 | 0 | 0
  Week 5, NCS, n=53, 50: number analyzed (Participants) | 53 | 50
  Week 5, NCS, n=53, 50 | 8 | 8
  Week 5, CS, n=53, 50: number analyzed (Participants) | 53 | 50
  Week 5, CS, n=53, 50 | 0 | 0
  Week 9, NCS, n=52, 46: number analyzed (Participants) | 52 | 46
  Week 9, NCS, n=52, 46 | 5 | 3
  Week 9, CS, n=52, 46: number analyzed (Participants) | 52 | 46
  Week 9, CS, n=52, 46 | 0 | 0
  Week 13, NCS, n=45, 40: number analyzed (Participants) | 45 | 40
  Week 13, NCS, n=45, 40 | 6 | 4
  Week 13, CS, n=45, 40: number analyzed (Participants) | 45 | 40
  Week 13, CS, n=45, 40 | 0 | 0
  Week 17, NCS, n=45, 36: number analyzed (Participants) | 45 | 36
  Week 17, NCS, n=45, 36 | 9 | 4
  Week 17, CS, n=45, 36: number analyzed (Participants) | 45 | 36
  Week 17, CS, n=45, 36 | 0 | 0
  Week 21, NCS, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, NCS, n=42, 34 | 3 | 1
  Week 21, CS, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, CS, n=42, 34 | 0 | 0
  Week 25, NCS, n=41, 31: number analyzed (Participants) | 41 | 31
  Week 25, NCS, n=41, 31 | 2 | 3
  Week 25, CS, n=41, 31: number analyzed (Participants) | 41 | 31
  Week 25, CS, n=41, 31 | 0 | 0

7. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters Including Blood Urea Nitrogen (BUN), Glucose Fasting, Chloride, Sodium, Potassium, Carbon Dioxide, and Calcium at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: BUN, glucose fasting, chloride, sodium, potassium, carbon dioxide (CO2), and calcium were assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Millimoles per liter (mmol/L)
  Calcium, Week 1, pre-dose, n=46, 46: number analyzed (Participants) | 46 | 46
  Calcium, Week 1, pre-dose, n=46, 46 | 2.33529 (0.07920) | 2.31724 (0.08132)
  Calcium, Week 2, n=53, 52 | 2.34262 (0.07908) | 2.35237 (0.09561)
  Calcium, Week 5, pre-dose, n=52, 49: number analyzed (Participants) | 52 | 49
  Calcium, Week 5, pre-dose, n=52, 49 | 2.31874 (0.09841) | 2.34182 (0.09948)
  Calcium, Week 9, pre-dose, n=52, 46: number analyzed (Participants) | 52 | 46
  Calcium, Week 9, pre-dose, n=52, 46 | 2.31885 (0.07624) | 2.36803 (0.18232)
  Calcium, Week 13, pre-dose, n=44, 40: number analyzed (Participants) | 44 | 40
  Calcium, Week 13, pre-dose, n=44, 40 | 2.32566 (0.07731) | 2.34848 (0.08552)
  Calcium, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Calcium, Week 17, pre-dose, n=45, 35 | 2.31207 (0.09495) | 2.35610 (0.10049)
  Calcium, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Calcium, Week 21, pre-dose, n=42, 34 | 2.30473 (0.08874) | 2.32699 (0.10993)
  Calcium, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  Calcium, Week 25, 4 weeks post last dose, n=41, 32 | 2.31374 (0.13942) | 2.36884 (0.08507)
  Chloride, Week 1, pre-dose, n=50, 51: number analyzed (Participants) | 50 | 51
  Chloride, Week 1, pre-dose, n=50, 51 | 103.7 (2.57) | 103.8 (2.52)
  Chloride, Week 2, n=50, 51: number analyzed (Participants) | 50 | 51
  Chloride, Week 2, n=50, 51 | 103.8 (2.23) | 103.5 (2.39)
  Chloride, Week 5, pre-dose, n=51, 49: number analyzed (Participants) | 51 | 49
  Chloride, Week 5, pre-dose, n=51, 49 | 103.5 (3.24) | 103.6 (2.34)
  Chloride, Week 9, pre-dose, n=51, 44: number analyzed (Participants) | 51 | 44
  Chloride, Week 9, pre-dose, n=51, 44 | 103.7 (2.85) | 103.6 (2.33)
  Chloride, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Chloride, Week 13, pre-dose, n=45, 40 | 103.4 (2.36) | 103.2 (2.55)
  Chloride, Week 17, pre-dose, n=45, 34: number analyzed (Participants) | 45 | 34
  Chloride, Week 17, pre-dose, n=45, 34 | 103.6 (2.72) | 103.4 (2.32)
  Chloride, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Chloride, Week 21, pre-dose, n=42, 34 | 103.6 (2.55) | 103.4 (2.53)
  Chloride, Week 25, 4 weeks post last dose, n=40,32: number analyzed (Participants) | 40 | 32
  Chloride, Week 25, 4 weeks post last dose, n=40,32 | 103.0 (2.36) | 103.2 (2.73)
  CO2, Week 1, pre-dose, n=47, 51: number analyzed (Participants) | 47 | 51
  CO2, Week 1, pre-dose, n=47, 51 | 27.3 (2.38) | 26.4 (2.31)
  CO2, Week 2, n=50, 50: number analyzed (Participants) | 50 | 50
  CO2, Week 2, n=50, 50 | 26.5 (2.71) | 26.4 (2.36)
  CO2, Week 5, pre-dose, n=50, 50: number analyzed (Participants) | 50 | 50
  CO2, Week 5, pre-dose, n=50, 50 | 26.4 (2.76) | 26.1 (2.66)
  CO2, Week 9, pre-dose, n=51, 45: number analyzed (Participants) | 51 | 45
  CO2, Week 9, pre-dose, n=51, 45 | 27.2 (2.63) | 26.1 (2.81)
  CO2, Week 13, pre-dose, n=45, 38: number analyzed (Participants) | 45 | 38
  CO2, Week 13, pre-dose, n=45, 38 | 27.4 (2.32) | 26.4 (2.11)
  CO2, Week 17, pre-dose, n=45, 34: number analyzed (Participants) | 45 | 34
  CO2, Week 17, pre-dose, n=45, 34 | 26.4 (2.98) | 26.3 (2.31)
  CO2, Week 21, pre-dose, n=40, 34: number analyzed (Participants) | 40 | 34
  CO2, Week 21, pre-dose, n=40, 34 | 27.2 (2.05) | 26.4 (2.39)
  CO2, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  CO2, Week 25, 4 weeks post last dose, n=41, 32 | 27.2 (2.73) | 27.0 (2.21)
  Glucose, Week 1, pre-dose, n=49, 51: number analyzed (Participants) | 49 | 51
  Glucose, Week 1, pre-dose, n=49, 51 | 5.02333 (1.06419) | 4.90943 (0.55713)
  Glucose, Week 2, n=49, 45: number analyzed (Participants) | 49 | 45
  Glucose, Week 2, n=49, 45 | 5.07525 (0.94855) | 4.85985 (0.69818)
  Glucose, Week 5, pre-dose, n=52, 49: number analyzed (Participants) | 52 | 49
  Glucose, Week 5, pre-dose, n=52, 49 | 4.97329 (0.75574) | 4.97545 (0.68857)
  Glucose, Week 9, pre-dose, n=50, 44: number analyzed (Participants) | 50 | 44
  Glucose, Week 9, pre-dose, n=50, 44 | 5.07978 (0.82661) | 5.01449 (0.70049)
  Glucose, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Glucose, Week 13, pre-dose, n=45, 40 | 5.09957 (0.90555) | 4.95848 (0.63337)
  Glucose, Week 17, pre-dose, n=44, 34: number analyzed (Participants) | 44 | 34
  Glucose, Week 17, pre-dose, n=44, 34 | 5.19291 (1.20604) | 4.99349 (0.65387)
  Glucose, Week 21, pre-dose, n=40, 33: number analyzed (Participants) | 40 | 33
  Glucose, Week 21, pre-dose, n=40, 33 | 5.12557 (1.14974) | 5.01559 (0.55765)
  Glucose, Week 25, 4 weeks post last dose, n=40, 31: number analyzed (Participants) | 40 | 31
  Glucose, Week 25, 4 weeks post last dose, n=40, 31 | 5.31222 (1.55173) | 5.08589 (0.57875)
  Potassium, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Potassium, Week 1, pre-dose, n=52, 52 | 4.11 (0.352) | 4.17 (0.353)
  Potassium, Week 2, n=53, 51: number analyzed (Participants) | 53 | 51
  Potassium, Week 2, n=53, 51 | 4.26 (0.345) | 4.23 (0.312)
  Potassium, Week 5, pre-dose, n=51, 49: number analyzed (Participants) | 51 | 49
  Potassium, Week 5, pre-dose, n=51, 49 | 4.10 (0.420) | 4.15 (0.357)
  Potassium, Week 9, pre-dose, n=52, 45: number analyzed (Participants) | 52 | 45
  Potassium, Week 9, pre-dose, n=52, 45 | 4.13 (0.364) | 4.19 (0.432)
  Potassium, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Potassium, Week 13, pre-dose, n=45, 40 | 4.09 (0.325) | 4.19 (0.378)
  Potassium, Week 17, pre-dose, n=44, 35: number analyzed (Participants) | 44 | 35
  Potassium, Week 17, pre-dose, n=44, 35 | 4.15 (0.389) | 4.28 (0.438)
  Potassium, Week 21, pre-dose, n=40, 34: number analyzed (Participants) | 40 | 34
  Potassium, Week 21, pre-dose, n=40, 34 | 4.19 (0.428) | 4.27 (0.415)
  Potassium, Week 25,4 weeks post last dose, n=41,32: number analyzed (Participants) | 41 | 32
  Potassium, Week 25,4 weeks post last dose, n=41,32 | 4.19 (0.404) | 4.29 (0.376)
  Sodium, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Sodium, Week 1, pre-dose, n=52, 52 | 141.9 (2.15) | 141.7 (2.15)
  Sodium, Week 2, n=53, 51: number analyzed (Participants) | 53 | 51
  Sodium, Week 2, n=53, 51 | 142.1 (1.95) | 141.5 (2.25)
  Sodium, Week 5, pre-dose, n=52, 49: number analyzed (Participants) | 52 | 49
  Sodium, Week 5, pre-dose, n=52, 49 | 141.7 (2.16) | 141.7 (1.91)
  Sodium, Week 9, pre-dose, n=52, 46: number analyzed (Participants) | 52 | 46
  Sodium, Week 9, pre-dose, n=52, 46 | 142.0 (2.27) | 141.5 (2.30)
  Sodium, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Sodium, Week 13, pre-dose, n=45, 40 | 141.8 (1.93) | 141.4 (2.47)
  Sodium, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Sodium, Week 17, pre-dose, n=45, 35 | 141.6 (2.34) | 141.5 (2.15)
  Sodium, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Sodium, Week 21, pre-dose, n=42, 34 | 141.5 (2.04) | 141.6 (2.48)
  Sodium, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  Sodium, Week 25, 4 weeks post last dose, n=41, 32 | 141.4 (2.11) | 141.7 (2.36)
  Urea, Week 1, pre-dose, n=51, 51: number analyzed (Participants) | 51 | 51
  Urea, Week 1, pre-dose, n=51, 51 | 7.6929 (3.69770) | 7.1568 (3.35084)
  Urea, Week 2, n=52, 52: number analyzed (Participants) | 52 | 52
  Urea, Week 2, n=52, 52 | 7.8847 (3.86054) | 7.1870 (3.81593)
  Urea, Week 5, pre-dose, n=52, 49: number analyzed (Participants) | 52 | 49
  Urea, Week 5, pre-dose, n=52, 49 | 7.9122 (3.86267) | 7.2488 (4.02159)
  Urea, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Urea, Week 9, pre-dose, n=51, 46 | 7.5806 (3.77958) | 7.0658 (3.40683)
  Urea, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Urea, Week 13, pre-dose, n=45, 40 | 7.4124 (3.50688) | 7.5311 (3.68104)
  Urea, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Urea, Week 17, pre-dose, n=45, 35 | 7.3499 (3.61940) | 7.9377 (3.59500)
  Urea, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Urea, Week 21, pre-dose, n=42, 34 | 7.7361 (3.58351) | 7.2357 (3.21507)
  Urea, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  Urea, Week 25, 4 weeks post last dose, n=41, 32 | 7.8770 (3.86299) | 6.9864 (3.01889)

8. Secondary Outcome: Absolute Values of the Clinical Chemistry Parameters of Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP), and Gamma Glutamyltransferase (GGT) at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: ALT, AST, ALP, and GGT were assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
International units per liter (IU/L)
  ALP, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  ALP, Week 1, pre-dose, n=52, 52 | 76.0 (17.09) | 67.8 (20.00)
  ALP, Week 2, n=53, 52 | 75.3 (15.92) | 69.0 (20.91)
  ALP, Week 5, pre-dose, n=51, 50: number analyzed (Participants) | 51 | 50
  ALP, Week 5, pre-dose, n=51, 50 | 75.1 (17.31) | 68.5 (21.84)
  ALP, Week 9, pre-dose, n=51, 45: number analyzed (Participants) | 51 | 45
  ALP, Week 9, pre-dose, n=51, 45 | 75.9 (17.63) | 69.8 (20.88)
  ALP, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  ALP, Week 13, pre-dose, n=45, 40 | 75.1 (16.92) | 69.7 (21.27)
  ALP, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  ALP, Week 17, pre-dose, n=45, 35 | 72.5 (16.30) | 69.5 (19.58)
  ALP, Week 21, pre-dose, n=41, 34: number analyzed (Participants) | 41 | 34
  ALP, Week 21, pre-dose, n=41, 34 | 72.4 (14.75) | 70.4 (21.81)
  ALP, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  ALP, Week 25, 4 weeks post last dose, n=41, 32 | 73.9 (14.56) | 72.4 (22.05)
  ALT, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  ALT, Week 1, pre-dose, n=52, 52 | 27.5 (13.33) | 26.1 (14.85)
  ALT, Week 2, n=53, 51: number analyzed (Participants) | 53 | 51
  ALT, Week 2, n=53, 51 | 26.3 (11.60) | 26.9 (15.89)
  ALT, Week 5, pre-dose, n=51, 50: number analyzed (Participants) | 51 | 50
  ALT, Week 5, pre-dose, n=51, 50 | 26.5 (15.11) | 25.0 (13.36)
  ALT, Week 9, pre-dose, n=52, 45: number analyzed (Participants) | 52 | 45
  ALT, Week 9, pre-dose, n=52, 45 | 26.4 (10.78) | 24.7 (12.41)
  ALT, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  ALT, Week 13, pre-dose, n=45, 40 | 29.1 (18.21) | 25.2 (11.18)
  ALT, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  ALT, Week 17, pre-dose, n=45, 35 | 25.7 (11.98) | 27.1 (15.11)
  ALT, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  ALT, Week 21, pre-dose, n=42, 34 | 26.2 (14.32) | 27.6 (14.02)
  ALT, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  ALT, Week 25, 4 weeks post last dose, n=41, 32 | 28.4 (15.43) | 26.4 (13.18)
  AST, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  AST, Week 1, pre-dose, n=52, 52 | 24.6 (7.73) | 25.5 (9.13)
  AST, Week 2, n=51, 51: number analyzed (Participants) | 51 | 51
  AST, Week 2, n=51, 51 | 24.2 (5.54) | 24.3 (7.51)
  AST, Week 5, pre-dose, n=51, 50: number analyzed (Participants) | 51 | 50
  AST, Week 5, pre-dose, n=51, 50 | 24.3 (6.51) | 23.6 (6.61)
  AST, Week 9, pre-dose, n=51, 45: number analyzed (Participants) | 51 | 45
  AST, Week 9, pre-dose, n=51, 45 | 24.6 (6.06) | 23.6 (5.94)
  AST, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  AST, Week 13, pre-dose, n=45, 40 | 25.4 (6.86) | 23.9 (6.04)
  AST, Week 17, pre-dose, n=44, 34: number analyzed (Participants) | 44 | 34
  AST, Week 17, pre-dose, n=44, 34 | 24.0 (8.34) | 23.9 (6.42)
  AST, Week 21, pre-dose, n=40, 34: number analyzed (Participants) | 40 | 34
  AST, Week 21, pre-dose, n=40, 34 | 24.5 (6.20) | 23.8 (5.18)
  AST, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  AST, Week 25, 4 weeks post last dose, n=41, 32 | 25.1 (5.63) | 24.0 (7.77)
  GGT, Week 1, pre-dose, n=50, 51: number analyzed (Participants) | 50 | 51
  GGT, Week 1, pre-dose, n=50, 51 | 34.4 (49.18) | 26.6 (20.37)
  GGT, Week 2, n=53, 52 | 32.6 (46.31) | 28.3 (24.67)
  GGT, Week 5, pre-dose, n=50, 50: number analyzed (Participants) | 50 | 50
  GGT, Week 5, pre-dose, n=50, 50 | 33.9 (59.91) | 28.0 (25.08)
  GGT, Week 9, pre-dose, n=50, 44: number analyzed (Participants) | 50 | 44
  GGT, Week 9, pre-dose, n=50, 44 | 33.7 (41.07) | 29.5 (24.86)
  GGT, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  GGT, Week 13, pre-dose, n=45, 40 | 37.2 (69.60) | 29.2 (21.56)
  GGT, Week 17, pre-dose, n=44,34: number analyzed (Participants) | 44 | 34
  GGT, Week 17, pre-dose, n=44,34 | 34.8 (57.83) | 34.6 (32.72)
  GGT, Week 21, pre-dose, n=41, 34: number analyzed (Participants) | 41 | 34
  GGT, Week 21, pre-dose, n=41, 34 | 38.6 (78.78) | 32.9 (27.27)
  GGT, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  GGT, Week 25, 4 weeks post last dose, n=41, 32 | 37.0 (54.09) | 28.4 (17.24)

9. Secondary Outcome: Absolute Values of the Clinical Chemistry Parameters of Albumin and Protein at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Albumin and protein were assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Grams per liter (g/L)
  Albumin, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Albumin, Week 1, pre-dose, n=52, 52 | 46.0 (3.00) | 46.1 (2.40)
  Albumin, Week 2, n=53, 52 | 45.2 (2.74) | 46.3 (3.17)
  Albumin, Week 5, pre-dose, n=52, 50: number analyzed (Participants) | 52 | 50
  Albumin, Week 5, pre-dose, n=52, 50 | 45.2 (2.46) | 45.8 (2.40)
  Albumin, Week 9, pre-dose, n=52, 46: number analyzed (Participants) | 52 | 46
  Albumin, Week 9, pre-dose, n=52, 46 | 45.3 (2.71) | 45.2 (2.51)
  Albumin, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Albumin, Week 13, pre-dose, n=45, 40 | 45.1 (2.26) | 45.8 (2.97)
  Albumin, Week 17, pre-dose, n=44, 35: number analyzed (Participants) | 44 | 35
  Albumin, Week 17, pre-dose, n=44, 35 | 44.8 (2.45) | 45.6 (2.13)
  Albumin, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Albumin, Week 21, pre-dose, n=42, 34 | 45.0 (2.69) | 45.1 (2.81)
  Albumin, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  Albumin, Week 25, 4 weeks post last dose, n=41, 32 | 45.7 (2.55) | 45.3 (2.50)
  Protein, Week 1, pre-dose, n=50, 48: number analyzed (Participants) | 50 | 48
  Protein, Week 1, pre-dose, n=50, 48 | 73.1 (5.09) | 73.7 (4.54)
  Protein, Week 2, n=52, 49: number analyzed (Participants) | 52 | 49
  Protein, Week 2, n=52, 49 | 72.4 (5.27) | 73.7 (5.30)
  Protein, Week 5, pre-dose, n=50, 49: number analyzed (Participants) | 50 | 49
  Protein, Week 5, pre-dose, n=50, 49 | 72.8 (5.33) | 72.6 (4.75)
  Protein, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Protein, Week 9, pre-dose, n=51, 46 | 73.0 (5.39) | 72.6 (4.50)
  Protein, Week 13, pre-dose, n=44, 40: number analyzed (Participants) | 44 | 40
  Protein, Week 13, pre-dose, n=44, 40 | 73.1 (4.76) | 72.8 (5.11)
  Protein, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Protein, Week 17, pre-dose, n=45, 35 | 71.3 (4.08) | 72.1 (4.26)
  Protein, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Protein, Week 21, pre-dose, n=42, 34 | 71.3 (4.30) | 71.4 (3.88)
  Protein, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  Protein, Week 25, 4 weeks post last dose, n=41, 32 | 72.1 (4.41) | 71.7 (4.53)

10. Secondary Outcome: Absolute Values of the Clinical Chemistry Parameters of Total and Direct Bilirubin, Creatinine (CRT), and Uric Acid (UA) at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Total bilirubin (TB) and direct bilirubin (DB), creatinine, and uric acid were assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Micromoles per liter
  UA, Week 1, pre-dose, n=48, 50: number analyzed (Participants) | 48 | 50
  UA, Week 1, pre-dose, n=48, 50 | 6280.75 (40503.47) | 9943.59 (47675.43)
  UA, Week 2, n=49, 49: number analyzed (Participants) | 49 | 49
  UA, Week 2, n=49, 49 | 7734.39 (50942.24) | 10906.56 (51211.16)
  UA, Week 5, pre-dose, n=50, 49: number analyzed (Participants) | 50 | 49
  UA, Week 5, pre-dose, n=50, 49 | 12991.02 (65048.95) | 13352.52 (64149.31)
  UA, Week 9, pre-dose, n=49, 44: number analyzed (Participants) | 49 | 44
  UA, Week 9, pre-dose, n=49, 44 | 13147.62 (62976.19) | 24031.30 (90312.49)
  UA, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  UA, Week 13, pre-dose, n=45, 40 | 14802.92 (69028.68) | 25208.07 (90067.04)
  UA, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  UA, Week 17, pre-dose, n=45, 35 | 15378.37 (70783.69) | 21723.77 (89724.11)
  UA, Week 21, pre-dose, n=40, 34: number analyzed (Participants) | 40 | 34
  UA, Week 21, pre-dose, n=40, 34 | 10414.21 (63827.10) | 22994.49 (94463.05)
  UA, Week 25, 4 weeks post last dose, n=40, 32: number analyzed (Participants) | 40 | 32
  UA, Week 25, 4 weeks post last dose, n=40, 32 | 9602.10 (58607.26) | 24506.63 (96050.66)
  CRT, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  CRT, Week 1, pre-dose, n=52, 52 | 80.2445 (15.71113) | 77.5162 (14.87768)
  CRT, Week 2, n=53, 51: number analyzed (Participants) | 53 | 51
  CRT, Week 2, n=53, 51 | 80.5450 (14.66619) | 78.3620 (13.55791)
  CRT, Week 5, pre-dose, n=52, 49: number analyzed (Participants) | 52 | 49
  CRT, Week 5, pre-dose, n=52, 49 | 79.0978 (14.80378) | 77.7282 (13.97357)
  CRT, Week 9, pre-dose, n=52, 46: number analyzed (Participants) | 52 | 46
  CRT, Week 9, pre-dose, n=52, 46 | 81.0171 (15.27077) | 75.9868 (13.78284)
  CRT, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  CRT, Week 13, pre-dose, n=45, 40 | 81.5454 (17.47683) | 77.5522 (13.18623)
  CRT, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  CRT, Week 17, pre-dose, n=45, 35 | 81.5074 (17.96973) | 76.7809 (12.15771)
  CRT, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  CRT, Week 21, pre-dose, n=42, 34 | 80.8093 (17.58041) | 75.1511 (11.77313)
  CRT, Week 25,4 weeks post last dose,n=41, 32: number analyzed (Participants) | 41 | 32
  CRT, Week 25,4 weeks post last dose,n=41, 32 | 81.9687 (17.48642) | 77.7839 (12.25219)
  TB, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  TB, Week 1, pre-dose, n=52, 52 | 9.878 (3.2705) | 10.595 (6.2074)
  TB, Week 2, n=53, 52 | 10.016 (4.5747) | 10.520 (4.1684)
  TB, Week 5, pre-dose, n=51, 50: number analyzed (Participants) | 51 | 50
  TB, Week 5, pre-dose, n=51, 50 | 10.189 (4.0635) | 10.878 (4.4865)
  TB, Week 9, pre-dose, n=51, 45: number analyzed (Participants) | 51 | 45
  TB, Week 9, pre-dose, n=51, 45 | 10.145 (3.5212) | 10.484 (4.2254)
  TB, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  TB, Week 13, pre-dose, n=45, 40 | 9.918 (3.6143) | 10.012 (5.0501)
  TB, Week 17, pre-dose, n=44, 35: number analyzed (Participants) | 44 | 35
  TB, Week 17, pre-dose, n=44, 35 | 10.624 (4.0522) | 9.877 (4.6822)
  TB, Week 21, pre-dose, n=40, 34: number analyzed (Participants) | 40 | 34
  TB, Week 21, pre-dose, n=40, 34 | 10.266 (3.6078) | 10.622 (6.0172)
  TB, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  TB, Week 25, 4 weeks post last dose, n=41, 32 | 9.820 (3.0792) | 10.162 (6.3294)
  DB, Week 1, pre-dose, n=50, 50: number analyzed (Participants) | 50 | 50
  DB, Week 1, pre-dose, n=50, 50 | 2.6685 (0.91566) | 2.8818 (1.54541)
  DB, Week 2, n=53, 51: number analyzed (Participants) | 53 | 51
  DB, Week 2, n=53, 51 | 2.9160 (1.02560) | 3.0690 (1.25759)
  DB, Week 5, pre-dose, n=49, 49: number analyzed (Participants) | 49 | 49
  DB, Week 5, pre-dose, n=49, 49 | 2.7981 (0.90148) | 2.9939 (1.12944)
  DB, Week 9, pre-dose, n=51, 43: number analyzed (Participants) | 51 | 43
  DB, Week 9, pre-dose, n=51, 43 | 2.9203 (1.10282) | 2.9693 (1.03703)
  DB, Week 13, pre-dose, n=43, 40: number analyzed (Participants) | 43 | 40
  DB, Week 13, pre-dose, n=43, 40 | 2.7958 (0.82254) | 3.0299 (1.55388)
  DB, Week 17, pre-dose, n=43, 35: number analyzed (Participants) | 43 | 35
  DB, Week 17, pre-dose, n=43, 35 | 2.9931 (0.85581) | 2.8714 (1.18421)
  DB, Week 21, pre-dose, n=39, 34: number analyzed (Participants) | 39 | 34
  DB, Week 21, pre-dose, n=39, 34 | 2.9267 (0.98861) | 3.0561 (1.33234)
  DB, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  DB, Week 25, 4 weeks post last dose, n=41, 32 | 3.0011 (0.95645) | 2.9864 (1.42919)

11. Secondary Outcome: Absolute Values of the Hematology Parameters of Platelet Count and White Blood Cell (WBC) Count, Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Platelet count, WBC count, basophils, eosinophils, lymphocytes, monocytes, and neutrophils were assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
10^9 cells per liter
  Platelets, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Platelets, Week 1, pre-dose, n=52, 52 | 246.1 (45.91) | 262.9 (53.61)
  Platelets, Week 2, n=53, 52 | 250.1 (47.25) | 264.6 (56.54)
  Platelets, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Platelets, Week 5, pre-dose, n=53, 50 | 240.7 (46.67) | 266.4 (61.20)
  Platelets, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Platelets, Week 9, pre-dose, n=51, 46 | 239.1 (43.29) | 267.0 (57.64)
  Platelets, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Platelets, Week 13, pre-dose, n=45, 40 | 242.7 (53.68) | 273.2 (56.18)
  Platelets, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Platelets, Week 17, pre-dose, n=45, 35 | 236.4 (45.59) | 270.2 (52.58)
  Platelets, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Platelets, Week 21, pre-dose, n=42, 34 | 233.0 (44.39) | 271.2 (53.89)
  Platelet, Week 25, 4 weeks post last dose, n=41,32: number analyzed (Participants) | 41 | 32
  Platelet, Week 25, 4 weeks post last dose, n=41,32 | 242.1 (48.64) | 279.3 (60.44)
  WBC, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  WBC, Week 1, pre-dose, n=52, 52 | 7.16 (1.794) | 6.81 (1.634)
  WBC, Week 2, n=53, 52 | 6.20 (1.535) | 6.90 (2.014)
  WBC, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  WBC, Week 5, pre-dose, n=53, 50 | 6.17 (1.580) | 6.77 (1.574)
  WBC, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  WBC, Week 9, pre-dose, n=51, 46 | 5.90 (1.508) | 6.92 (1.553)
  WBC, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  WBC, Week 13, pre-dose, n=45, 40 | 5.93 (1.541) | 7.18 (2.095)
  WBC, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  WBC, Week 17, pre-dose, n=45, 35 | 6.03 (1.780) | 6.99 (1.916)
  WBC, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  WBC, Week 21, pre-dose, n=42, 34 | 5.86 (1.143) | 6.92 (1.576)
  WBC, Week 25, 4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  WBC, Week 25, 4 weeks post last dose, n=41, 32 | 5.93 (1.357) | 7.00 (1.922)
  Basophils, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Basophils, Week 1, pre-dose, n=52, 52 | 0.05 (0.029) | 0.05 (0.026)
  Basophils, Week 2, n=53, 51: number analyzed (Participants) | 53 | 51
  Basophils, Week 2, n=53, 51 | 0.03 (0.021) | 0.05 (0.026)
  Basophils, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Basophils, Week 5, pre-dose, n=53, 50 | 0.02 (0.013) | 0.05 (0.032)
  Basophils, Week 9, pre-dose, n=51, 45: number analyzed (Participants) | 51 | 45
  Basophils, Week 9, pre-dose, n=51, 45 | 0.03 (0.017) | 0.05 (0.028)
  Basophils, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Basophils, Week 13, pre-dose, n=45, 40 | 0.03 (0.024) | 0.06 (0.082)
  Basophils, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Basophils, Week 17, pre-dose, n=45, 35 | 0.03 (0.021) | 0.05 (0.027)
  Basophils, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Basophils, Week 21, pre-dose, n=42, 34 | 0.03 (0.021) | 0.05 (0.041)
  Basophil, Week 25, 4 weeks post last dose, n=41,32: number analyzed (Participants) | 41 | 32
  Basophil, Week 25, 4 weeks post last dose, n=41,32 | 0.03 (0.021) | 0.05 (0.023)
  Eosinophils, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Eosinophils, Week 1, pre-dose, n=52, 52 | 0.63 (0.496) | 0.54 (0.305)
  Eosinophils, Week 2, n=53, 52 | 0.10 (0.079) | 0.55 (0.346)
  Eosinophils, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Eosinophils, Week 5, pre-dose, n=53, 50 | 0.05 (0.030) | 0.51 (0.276)
  Eosinophils, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Eosinophils, Week 9, pre-dose, n=51, 46 | 0.04 (0.027) | 0.55 (0.392)
  Eosinophils, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Eosinophils, Week 13, pre-dose, n=45, 40 | 0.07 (0.196) | 0.56 (0.476)
  Eosinophils, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Eosinophils, Week 17, pre-dose, n=45, 35 | 0.05 (0.125) | 0.45 (0.314)
  Eosinophils, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Eosinophils, Week 21, pre-dose, n=42, 34 | 0.04 (0.023) | 0.49 (0.411)
  Eosinophil, Week 25,4 weeks post last dose,n=41,32: number analyzed (Participants) | 41 | 32
  Eosinophil, Week 25,4 weeks post last dose,n=41,32 | 0.04 (0.029) | 0.44 (0.256)
  Lymphocytes, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Lymphocytes, Week 1, pre-dose, n=52, 52 | 1.94 (0.568) | 1.99 (0.615)
  Lymphocytes, Week 2, n=53, 52 | 1.84 (0.531) | 1.96 (0.516)
  Lymphocytes, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Lymphocytes, Week 5, pre-dose, n=53, 50 | 1.83 (0.635) | 1.90 (0.466)
  Lymphocytes, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Lymphocytes, Week 9, pre-dose, n=51, 46 | 1.83 (0.596) | 2.03 (0.616)
  Lymphocytes, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Lymphocytes, Week 13, pre-dose, n=45, 40 | 1.80 (0.457) | 2.02 (0.555)
  Lymphocytes, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Lymphocytes, Week 17, pre-dose, n=45, 35 | 1.77 (0.466) | 1.92 (0.453)
  Lymphocytes, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Lymphocytes, Week 21, pre-dose, n=42, 34 | 1.83 (0.541) | 1.98 (0.514)
  Lymphocyte,Week 25,4 weeks post last dose,n=41, 32: number analyzed (Participants) | 41 | 32
  Lymphocyte,Week 25,4 weeks post last dose,n=41, 32 | 1.88 (0.604) | 1.91 (0.523)
  Monocytes, Week 1, pre-dose, n=52, 51: number analyzed (Participants) | 52 | 51
  Monocytes, Week 1, pre-dose, n=52, 51 | 0.56 (0.166) | 0.50 (0.131)
  Monocytes, Week 2, n=53, 52 | 0.56 (0.175) | 0.54 (0.190)
  Monocytes, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Monocytes, Week 5, pre-dose, n=53, 50 | 0.53 (0.170) | 0.51 (0.138)
  Monocytes, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Monocytes, Week 9, pre-dose, n=51, 46 | 0.50 (0.140) | 0.53 (0.163)
  Monocytes, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Monocytes, Week 13, pre-dose, n=45, 40 | 0.50 (0.188) | 0.55 (0.159)
  Monocytes, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Monocytes, Week 17, pre-dose, n=45, 35 | 0.51 (0.172) | 0.52 (0.142)
  Monocytes, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Monocytes, Week 21, pre-dose, n=42, 34 | 0.50 (0.150) | 0.55 (0.158)
  Monocytes, Week 25,4 weeks post last dose,n=41, 32: number analyzed (Participants) | 41 | 32
  Monocytes, Week 25,4 weeks post last dose,n=41, 32 | 0.51 (0.130) | 0.57 (0.201)
  Neutrophils, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Neutrophils, Week 1, pre-dose, n=52, 52 | 3.96481 (1.374461) | 3.72673 (1.085727)
  Neutrophils, Week 2, n=53, 52 | 3.65642 (1.295348) | 3.80635 (1.525888)
  Neutrophils, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Neutrophils, Week 5, pre-dose, n=53, 50 | 3.73509 (1.238233) | 3.78720 (1.237163)
  Neutrophils, Week 9, pre-dose, n=51, 45: number analyzed (Participants) | 51 | 45
  Neutrophils, Week 9, pre-dose, n=51, 45 | 3.49333 (1.160355) | 3.76333 (1.095441)
  Neutrophils, Week 13, pre-dose, n=45, 39: number analyzed (Participants) | 45 | 39
  Neutrophils, Week 13, pre-dose, n=45, 39 | 3.52400 (1.287322) | 3.96169 (1.563461)
  Neutrophils, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Neutrophils, Week 17, pre-dose, n=45, 35 | 3.65711 (1.624295) | 4.06657 (1.550068)
  Neutrophils, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Neutrophils, Week 21, pre-dose, n=42, 34 | 3.45738 (0.907831) | 3.83824 (1.137039)
  Neutrophil,Week 25,4 weeks post last dose,n=41, 32: number analyzed (Participants) | 41 | 32
  Neutrophil,Week 25,4 weeks post last dose,n=41, 32 | 3.46854 (1.045869) | 4.03125 (1.452175)

12. Secondary Outcome: Absolute Values of the Hematology Parameters of Hemoglobin and Mean Corpuscular Hemoglobin Concentration (MCHC) at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Hemoglobin and MCHC were assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Grams per liter (g/L)
  Hemoglobin, Week 1, pre-dose, n=51, 52: number analyzed (Participants) | 51 | 52
  Hemoglobin, Week 1, pre-dose, n=51, 52 | 148.445 (11.5174) | 145.566 (22.1192)
  Hemoglobin, Week 2, n=53, 52 | 148.013 (12.2563) | 147.625 (11.1436)
  Hemoglobin, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Hemoglobin, Week 5, pre-dose, n=53, 50 | 147.955 (10.8860) | 146.071 (12.7175)
  Hemoglobin, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Hemoglobin, Week 9, pre-dose, n=51, 46 | 147.135 (11.0248) | 146.252 (12.0539)
  Hemoglobin, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Hemoglobin, Week 13, pre-dose, n=45, 40 | 147.498 (10.9510) | 147.427 (11.9305)
  Hemoglobin, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Hemoglobin, Week 17, pre-dose, n=45, 35 | 145.988 (11.4327) | 148.045 (12.0595)
  Hemoglobin, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Hemoglobin, Week 21, pre-dose, n=42, 34 | 146.597 (11.8831) | 146.953 (10.9213)
  Hemoglobin,Week 25,4 weeks post last dose,n=41, 32: number analyzed (Participants) | 41 | 32
  Hemoglobin,Week 25,4 weeks post last dose,n=41, 32 | 148.927 (10.5835) | 147.940 (8.9890)
  MCHC, Week 1, pre-dose, n=52, 51: number analyzed (Participants) | 52 | 51
  MCHC, Week 1, pre-dose, n=52, 51 | 338.3 (8.71) | 338.6 (16.71)
  MCHC, Week 2, n=52, 52: number analyzed (Participants) | 52 | 52
  MCHC, Week 2, n=52, 52 | 338.1 (10.34) | 335.2 (9.33)
  MCHC, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  MCHC, Week 5, pre-dose, n=53, 50 | 338.1 (7.71) | 338.6 (15.85)
  MCHC, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  MCHC, Week 9, pre-dose, n=51, 46 | 336.5 (10.40) | 337.7 (9.52)
  MCHC, Week 13, pre-dose, n=44, 40: number analyzed (Participants) | 44 | 40
  MCHC, Week 13, pre-dose, n=44, 40 | 338.7 (9.52) | 339.6 (17.77)
  MCHC, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  MCHC, Week 17, pre-dose, n=45, 35 | 338.6 (9.56) | 337.0 (10.02)
  MCHC, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  MCHC, Week 21, pre-dose, n=42, 34 | 338.9 (9.35) | 336.4 (9.84)
  MCHC, Week 25,4 weeks post last dose,n=40, 32: number analyzed (Participants) | 40 | 32
  MCHC, Week 25,4 weeks post last dose,n=40, 32 | 338.9 (9.23) | 339.3 (18.86)

13. Secondary Outcome: Absolute Values of the Hematology Parameter of Red Blood Cell (RBC) Count and Reticulocyte Count (RC) at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: RBC count and RC were assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10^12 cells per litre
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
10^12 cells per litre
  RBC, Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  RBC, Week 1, pre-dose, n=52, 52 | 4.889 (0.3758) | 4.930 (0.4830)
  RBC, Week 2, n=53, 52 | 4.868 (0.4024) | 4.937 (0.4340)
  RBC, Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  RBC, Week 5, pre-dose, n=53, 50 | 4.876 (0.3494) | 4.867 (0.5115)
  RBC, Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  RBC, Week 9, pre-dose, n=51, 46 | 4.875 (0.3792) | 4.879 (0.4758)
  RBC, Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  RBC, Week 13, pre-dose, n=45, 40 | 4.889 (0.3511) | 4.923 (0.4828)
  RBC, Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  RBC, Week 17, pre-dose, n=45, 35 | 4.824 (0.3735) | 4.938 (0.5058)
  RBC, Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  RBC, Week 21, pre-dose, n=42, 34 | 4.840 (0.3743) | 4.910 (0.5165)
  RBC, Week 25,4 weeks post last dose,n=41, 32: number analyzed (Participants) | 41 | 32
  RBC, Week 25,4 weeks post last dose,n=41, 32 | 4.902 (0.3551) | 4.901 (0.3343)
  RC, Week 1, pre-dose, n=28, 32: number analyzed (Participants) | 28 | 32
  RC, Week 1, pre-dose, n=28, 32 | 0.0537 (0.01651) | 0.0495 (0.01666)
  RC, Week 2, n=33, 35: number analyzed (Participants) | 33 | 35
  RC, Week 2, n=33, 35 | 0.0495 (0.01682) | 0.0506 (0.01879)
  RC, Week 5, pre-dose, n=33, 33: number analyzed (Participants) | 33 | 33
  RC, Week 5, pre-dose, n=33, 33 | 0.0461 (0.01416) | 0.0496 (0.02530)
  RC, Week 9, pre-dose, n=29, 29: number analyzed (Participants) | 29 | 29
  RC, Week 9, pre-dose, n=29, 29 | 0.0443 (0.01327) | 0.0513 (0.02581)
  RC, Week 13, pre-dose, n=28, 23: number analyzed (Participants) | 28 | 23
  RC, Week 13, pre-dose, n=28, 23 | 0.0473 (0.01530) | 0.0528 (0.01780)
  RC, Week 17, pre-dose, n=28, 20: number analyzed (Participants) | 28 | 20
  RC, Week 17, pre-dose, n=28, 20 | 0.0482 (0.01604) | 0.0493 (0.01847)
  RC, Week 21, pre-dose, n=26, 19: number analyzed (Participants) | 26 | 19
  RC, Week 21, pre-dose, n=26, 19 | 0.0459 (0.01592) | 0.0521 (0.01594)
  RC, Week 25,4 weeks post last dose,n=24, 20: number analyzed (Participants) | 24 | 20
  RC, Week 25,4 weeks post last dose,n=24, 20 | 0.0489 (0.01640) | 0.0580 (0.02625)

14. Secondary Outcome: Absolute Values of the Hematology Parameter of Mean Corpuscular Hemoglobin (MCH) at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: MCH was assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Picograms (pg)
  Week 1, pre-dose, n=52, 51: number analyzed (Participants) | 52 | 51
  Week 1, pre-dose, n=52, 51 | 30.44 (1.215) | 30.26 (1.804)
  Week 2, n=52, 52: number analyzed (Participants) | 52 | 52
  Week 2, n=52, 52 | 30.46 (1.359) | 29.94 (1.631)
  Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Week 5, pre-dose, n=53, 50 | 30.37 (1.301) | 30.10 (1.686)
  Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Week 9, pre-dose, n=51, 46 | 30.23 (1.378) | 30.07 (1.793)
  Week 13, pre-dose, n=44, 40: number analyzed (Participants) | 44 | 40
  Week 13, pre-dose, n=44, 40 | 30.22 (1.292) | 29.94 (2.187)
  Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Week 17, pre-dose, n=45, 35 | 30.29 (1.339) | 30.10 (1.951)
  Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, pre-dose, n=42, 34 | 30.33 (1.354) | 30.00 (2.035)
  Week 25,4 weeks post last dose,n=40, 32: number analyzed (Participants) | 40 | 32
  Week 25,4 weeks post last dose,n=40, 32 | 30.41 (1.196) | 30.26 (1.243)

15. Secondary Outcome: Absolute Values of the Hematology Parameter of Mean Corpuscular Volume (MCV) at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: MCV was assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Femtoliters
  Week 1, pre-dose, n=52, 52: number analyzed (Participants) | 52 | 52
  Week 1, pre-dose, n=52, 52 | 90.04 (3.850) | 89.43 (5.051)
  Week 2, n=53, 52 | 90.06 (3.997) | 89.41 (4.765)
  Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Week 5, pre-dose, n=53, 50 | 89.85 (3.911) | 89.38 (4.876)
  Week 9, pre-dose, n=51, 46: number analyzed (Participants) | 51 | 46
  Week 9, pre-dose, n=51, 46 | 89.81 (3.897) | 89.07 (5.019)
  Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Week 13, pre-dose, n=45, 40 | 89.19 (3.934) | 89.12 (5.358)
  Week 17, pre-dose, n=45, 35: number analyzed (Participants) | 45 | 35
  Week 17, pre-dose, n=45, 35 | 89.50 (3.714) | 89.33 (5.469)
  Week 21, pre-dose, n=42, 34: number analyzed (Participants) | 42 | 34
  Week 21, pre-dose, n=42, 34 | 89.46 (3.673) | 89.23 (5.542)
  Week 25,4 weeks post last dose, n=41, 32: number analyzed (Participants) | 41 | 32
  Week 25,4 weeks post last dose, n=41, 32 | 89.68 (3.364) | 89.91 (3.831)

16. Secondary Outcome: Absolute Value of the Hematology Parameter of Reticulocyte Count/Erythrocyte Uncorrected at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Reticulocyte count was assessed at Week 1 pre-dose, Week 2, Week 5 pre-dose, Week 9 pre-dose, Week 13 pre-dose, Week 17 pre-dose, Week 21 pre-dose, and Week 25 (4 Weeks post last dose).
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 19 | 16
Ratio
  Week 1, pre-dose, n=19, 16 | 0.1723 (0.16091) | 0.1053 (0.05750)
  Week 2, n=19, 16 | 0.1710 (0.15032) | 0.1271 (0.09305)
  Week 5, pre-dose, n=19, 16 | 0.1731 (0.16016) | 0.1464 (0.13471)
  Week 9, pre-dose, n=18, 16: number analyzed (Participants) | 18 | 16
  Week 9, pre-dose, n=18, 16 | 0.1556 (0.12224) | 0.1299 (0.10015)
  Week 13, pre-dose, n=15, 16: number analyzed (Participants) | 15 | 16
  Week 13, pre-dose, n=15, 16 | 0.1483 (0.12563) | 0.1324 (0.10103)
  Week 17, pre-dose, n=15, 14: number analyzed (Participants) | 15 | 14
  Week 17, pre-dose, n=15, 14 | 0.1645 (0.17438) | 0.1423 (0.13603)
  Week 21, pre-dose, n=15, 13: number analyzed (Participants) | 15 | 13
  Week 21, pre-dose, n=15, 13 | 0.1446 (0.11350) | 0.1395 (0.11754)
  Week 25,4 weeks post last dose, n=15, 12: number analyzed (Participants) | 15 | 12
  Week 25,4 weeks post last dose, n=15, 12 | 0.1465 (0.12045) | 0.1402 (0.09660)

17. Secondary Outcome: Number of Participants With Positive Clinically Relevant Urinalysis Results at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Specific gravity, power of hydrogen (pH), glucose, protein, blood, and ketones were assessed at Weeks (Wk) 1, 2, 5, 9, 13, 17, 21, and 25. Results for all urinalysis parameters were assessed for clinical relevance by physician. Clinically relevant positive results are presented. Clinically relevant positive results are defined as those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Clinically relevant positive results Wk 1, n=53,52 | 0 | 0
  Clinically relevant positive results Wk 2, n=46,49: number analyzed (Participants) | 46 | 49
  Clinically relevant positive results Wk 2, n=46,49 | 0 | 0
  Clinically relevant positive results Wk 5, n=53,50: number analyzed (Participants) | 53 | 50
  Clinically relevant positive results Wk 5, n=53,50 | 0 | 0
  Clinically relevant positive results Wk 9, n=51,46: number analyzed (Participants) | 51 | 46
  Clinically relevant positive results Wk 9, n=51,46 | 0 | 0
  Clinically relevant positive results Wk 13,n=45,40: number analyzed (Participants) | 45 | 40
  Clinically relevant positive results Wk 13,n=45,40 | 0 | 0
  Clinically relevant positive results Wk 17,n=45,36: number analyzed (Participants) | 45 | 36
  Clinically relevant positive results Wk 17,n=45,36 | 0 | 0
  Clinically relevant positive results Wk 21,n=42,34: number analyzed (Participants) | 42 | 34
  Clinically relevant positive results Wk 21,n=42,34 | 0 | 0
  Clinically relevant positive results Wk 25,n=39,31: number analyzed (Participants) | 39 | 31
  Clinically relevant positive results Wk 25,n=39,31 | 0 | 0

18. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is an important medical event that jeopardizes the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or is associated with liver injury and impaired liver function.
Time Frame: Up to 11 months
Population: Safety Population. One participant randomized to mepolizumab took placebo in error. Thus, "N" for the placebo arm of the SP is greater than for the ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Any AE | 40 | 42
  Any SAE | 0 | 0

19. Secondary Outcome: Mean of the Forced Expiratory Volume in 1 Second (FEV1) at Weeks 2, 5, 9, 13, 17, 21, and 25
Description: FEV1 is defined as the volume of air forcefully expelled from the lungs in one second. FEV1 measurements were taken by spirometry at each clinic visit. FEV1 was calculated as the maximum of three readings taken at each time point for each participant. Spirometry data is plotted and analyzed using a repeated measures model to calculate treatment difference, confidence intervals and p-values.
Time Frame: Weeks 2, 5, 9, 13, 17, 21, and 25
Population: ITT Population: all randomized participants who received at least one dose of study treatment. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters (L)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
Liters (L)
  Week 2, n=54, 51 | 3.24 [3.14 to 3.35] | 3.20 [3.10 to 3.31]
  Week 5, n=54, 49: number analyzed (Participants) | 54 | 49
  Week 5, n=54, 49 | 3.33 [3.23 to 3.44] | 3.28 [3.17 to 3.39]
  Week 9, n=47, 44: number analyzed (Participants) | 47 | 44
  Week 9, n=47, 44 | 3.32 [3.19 to 3.45] | 3.23 [3.09 to 3.37]
  Week 13, n=44, 37: number analyzed (Participants) | 44 | 37
  Week 13, n=44, 37 | 3.35 [3.23 to 3.47] | 3.18 [3.06 to 3.31]
  Week 17, n=43, 34: number analyzed (Participants) | 43 | 34
  Week 17, n=43, 34 | 3.33 [3.18 to 3.48] | 3.12 [2.96 to 3.28]
  Week 21, n=42, 32: number analyzed (Participants) | 42 | 32
  Week 21, n=42, 32 | 3.41 [3.27 to 3.54] | 3.18 [3.04 to 3.33]
  Week 25, n=42, 32: number analyzed (Participants) | 42 | 32
  Week 25, n=42, 32 | 3.35 [3.23 to 3.47] | 3.18 [3.05 to 3.32]
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.567, repeated measures model; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.10 to 0.19] — Week 2
Statistical Analysis 2: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.495, repeated measures model; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.10 to 0.21] — Week 5
Statistical Analysis 3: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.365, repeated measures model; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.10 to 0.28] — Week 9
Statistical Analysis 4: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.058, repeated measures model; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.01 to 0.34] — Week 13
Statistical Analysis 5: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.056, repeated measures model; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.01 to 0.43] — Week 17
Statistical Analysis 6: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.028, repeated measures model; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [0.03 to 0.42] — Week 21
Statistical Analysis 7: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.077, repeated measures model; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.02 to 0.34] — Week 25

20. Secondary Outcome: Mean of Forced Vital Capacity (FVC) at Weeks 2, 5, 9, 13, 17, 21, and 25
Description: FVC is defined as the maximum amount of air that can forcibly be blown out after a maximum inspiration. FVC was calculated as the maximum of three readings taken at each time point for each participant. Spirometry data are plotted and analyzed using a repeated measures model to calculate treatment difference, confidence intervals and p-values.
Time Frame: Weeks 2, 5, 9, 13, 17, 21, and 25
Population: ITT Population. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
Liters
  Week 2, n=54, 51 | 4.51 [4.39 to 4.62] | 4.45 [4.34 to 4.56]
  Week 5, n=54, 49: number analyzed (Participants) | 54 | 49
  Week 5, n=54, 49 | 4.55 [4.45 to 4.66] | 4.49 [4.38 to 4.60]
  Week 9, n=47, 44: number analyzed (Participants) | 47 | 44
  Week 9, n=47, 44 | 4.52 [4.38 to 4.66] | 4.46 [4.32 to 4.60]
  Week 13, n=44, 37: number analyzed (Participants) | 44 | 37
  Week 13, n=44, 37 | 4.62 [4.49 to 4.75] | 4.43 [4.28 to 4.57]
  Week 17, n=43, 34: number analyzed (Participants) | 43 | 34
  Week 17, n=43, 34 | 4.59 [4.43 to 4.74] | 4.37 [4.19 to 4.54]
  Week 21, n=42, 32: number analyzed (Participants) | 42 | 32
  Week 21, n=42, 32 | 4.66 [4.51 to 4.81] | 4.38 [4.22 to 4.55]
  Week 25, n=42, 32: number analyzed (Participants) | 42 | 32
  Week 25, n=42, 32 | 4.59 [4.45 to 4.74] | 4.41 [4.25 to 4.57]
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.486, repeated measures model; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.10 to 0.22] — Week 2
Statistical Analysis 2: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.384, repeated measures model; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.08 to 0.22] — Week 5
Statistical Analysis 3: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.546, repeated measures model; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.14 to 0.26] — Week 9
Statistical Analysis 4: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.050, repeated measures model; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [0.00 to 0.39] — Week 13
Statistical Analysis 5: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.061, repeated measures model; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.01 to 0.45] — Week 17
Statistical Analysis 6: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.016, repeated measures model; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.05 to 0.51] — Week 21
Statistical Analysis 7: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.094, repeated measures model; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.03 to 0.40] — Week 25

21. Secondary Outcome: Mean Peak Expiratory Flow Rate (PEFR) at Indicated Weeks 2, 5, 9, 13, 17, 21, and 25
Description: PEFR is defined as the maximum airflowrate generated during a forced expiration beginning with the lungs fully inflated. PEFR was calculated as the maximum of three readings taken at each time point for each participant. Spirometry data is plotted and analyzed using a repeated measures model to calculate treatment difference, confidence intervals and p-values.
Time Frame: Weeks 2, 5, 9, 13, 17, 21, and 25
Population: ITT Population. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/minute (L/min)
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
Liters/minute (L/min)
  Week 2, n=54, 51 | 472.81 [455.37 to 490.25] | 467.70 [449.78 to 485.63]
  Week 5, n=54, 49: number analyzed (Participants) | 54 | 49
  Week 5, n=54, 49 | 489.08 [469.08 to 509.07] | 474.53 [453.61 to 495.45]
  Week 9, n=47, 45: number analyzed (Participants) | 47 | 45
  Week 9, n=47, 45 | 487.07 [462.19 to 511.95] | 478.16 [452.57 to 503.75]
  Week 13, n=44, 37: number analyzed (Participants) | 44 | 37
  Week 13, n=44, 37 | 494.04 [470.85 to 517.23] | 470.81 [445.97 to 495.65]
  Week 17, n=43, 34: number analyzed (Participants) | 43 | 34
  Week 17, n=43, 34 | 493.68 [467.67 to 519.69] | 455.52 [427.15 to 483.89]
  Week 21, n=42, 32: number analyzed (Participants) | 42 | 32
  Week 21, n=42, 32 | 501.88 [476.83 to 526.93] | 463.17 [435.53 to 490.81]
  Week 25, n=42, 32: number analyzed (Participants) | 42 | 32
  Week 25, n=42, 32 | 481.05 [454.31 to 507.79] | 466.93 [437.33 to 496.52]
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.686, repeated measures model; Mean Difference (Final Values) = 5.11, 95% CI 2-sided [-19.91 to 30.12] — Week 2
Statistical Analysis 2: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.321, repeated measures model; Mean Difference (Final Values) = 14.55, 95% CI 2-sided [-14.40 to 43.50] — Week 5
Statistical Analysis 3: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.622, repeated measures model; Mean Difference (Final Values) = 8.91, 95% CI 2-sided [-26.79 to 44.60] — Week 9
Statistical Analysis 4: Comparison: Mepolizumab 750 mg; Test type: Superiority or Other; p = 0.178, repeated measures model; Mean Difference (Final Values) = 23.24, 95% CI 2-sided [-10.75 to 57.22] — Week 13
Statistical Analysis 5: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.052, repeated measures model; Mean Difference (Final Values) = 38.16, 95% CI 2-sided [-0.33 to 76.66] — Week 17
Statistical Analysis 6: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.042, repeated measures model; Mean Difference (Final Values) = 38.72, 95% CI 2-sided [1.41 to 76.02] — Week 21
Statistical Analysis 7: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.484, repeated measures model; Mean Difference (Final Values) = 14.13, 95% CI 2-sided [-25.76 to 54.02] — Week 25

22. Secondary Outcome: Individual Symptoms Visual Analogue Scale (VAS) Scores at Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Description: Participants were asked to indicate on a VAS (0 to 10 centimeters) the severity of nasal polyposis and its four symptoms (one VAS for each symptom): rhinorrhea; mucus in the throat; nasal blockage; loss of smell. The left-hand side of the scale (0) represents "not troublesome," and the right hand side of the scale (10) represents "worst possible troublesome." Hence the score ranges between 0 to 10, with higher scores indicating greater severity.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21, and 25
Population: PP Population. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 49 | 51
Scores on a scale
  Nasal Polyposis, Week 1, n=49, 51 | 8.51 (0.928) | 8.64 (1.101)
  Nasal Polyposis, Week 2, n=49, 51 | 7.91 (1.766) | 8.47 (1.326)
  Nasal Polyposis, Week 5, n=49, 49: number analyzed (Participants) | 49 | 49
  Nasal Polyposis, Week 5, n=49, 49 | 7.10 (2.310) | 7.75 (2.083)
  Nasal Polyposis, Week 9, n=47, 46: number analyzed (Participants) | 47 | 46
  Nasal Polyposis, Week 9, n=47, 46 | 6.14 (3.022) | 7.74 (2.112)
  Nasal Polyposis, Week 13, n=45, 39: number analyzed (Participants) | 45 | 39
  Nasal Polyposis, Week 13, n=45, 39 | 5.79 (3.524) | 7.21 (2.563)
  Nasal Polyposis, Week 17, n=44, 34: number analyzed (Participants) | 44 | 34
  Nasal Polyposis, Week 17, n=44, 34 | 5.00 (3.518) | 6.44 (3.164)
  Nasal Polyposis, Week 21, n=42, 33: number analyzed (Participants) | 42 | 33
  Nasal Polyposis, Week 21, n=42, 33 | 4.70 (3.513) | 6.47 (3.098)
  Nasal Polyposis, Week 25, n=42, 31: number analyzed (Participants) | 42 | 31
  Nasal Polyposis, Week 25, n=42, 31 | 4.16 (3.582) | 6.21 (3.357)
  Rhinorrhea, Week 1, n=49, 51 | 6.60 (2.694) | 6.17 (3.086)
  Rhinorrhea, Week 2, n=49, 51 | 5.59 (2.863) | 6.28 (2.992)
  Rhinorrhea, Week 5, n=49, 49: number analyzed (Participants) | 49 | 49
  Rhinorrhea, Week 5, n=49, 49 | 4.98 (3.365) | 5.98 (2.926)
  Rhinorrhea, Week 9, n=48, 46: number analyzed (Participants) | 48 | 46
  Rhinorrhea, Week 9, n=48, 46 | 4.65 (3.309) | 6.28 (3.129)
  Rhinorrhea, Week 13, n=45, 39: number analyzed (Participants) | 45 | 39
  Rhinorrhea, Week 13, n=45, 39 | 4.18 (3.340) | 5.19 (3.106)
  Rhinorrhea, Week 17, n=44, 34: number analyzed (Participants) | 44 | 34
  Rhinorrhea, Week 17, n=44, 34 | 3.33 (3.338) | 4.82 (3.399)
  Rhinorrhea, Week 21, n=42, 34: number analyzed (Participants) | 42 | 34
  Rhinorrhea, Week 21, n=42, 34 | 3.50 (3.408) | 4.70 (3.512)
  Rhinorrhea, Week 25, n=42, 31: number analyzed (Participants) | 42 | 31
  Rhinorrhea, Week 25, n=42, 31 | 3.03 (3.428) | 4.71 (3.812)
  Mucus in Throat, Week 1, n=49, 51 | 5.92 (2.878) | 6.53 (2.732)
  Mucus in Throat, Week 2, n=49, 51 | 5.27 (2.807) | 6.15 (2.764)
  Mucus in Throat, Week 5, n=49, 49: number analyzed (Participants) | 49 | 49
  Mucus in Throat, Week 5, n=49, 49 | 4.92 (3.012) | 5.92 (2.640)
  Mucus in Throat, Week 9, n=48, 46: number analyzed (Participants) | 48 | 46
  Mucus in Throat, Week 9, n=48, 46 | 3.93 (3.232) | 6.37 (2.942)
  Mucus in Throat, Week 13, n=45, 39: number analyzed (Participants) | 45 | 39
  Mucus in Throat, Week 13, n=45, 39 | 4.11 (3.079) | 5.49 (3.280)
  Mucus in Throat, Week 17, n=44, 34: number analyzed (Participants) | 44 | 34
  Mucus in Throat, Week 17, n=44, 34 | 3.28 (3.190) | 5.16 (3.482)
  Mucus in Throat, Week 21, n=42, 34: number analyzed (Participants) | 42 | 34
  Mucus in Throat, Week 21, n=42, 34 | 3.30 (3.356) | 4.84 (3.457)
  Mucus in Throat, Week 25, n=42, 31: number analyzed (Participants) | 42 | 31
  Mucus in Throat, Week 25, n=42, 31 | 3.24 (3.263) | 5.23 (3.405)
  Nasal Blockage, Week 1, n=49, 51 | 7.76 (2.459) | 8.36 (1.783)
  Nasal Blockage, Week 2, n=49, 51 | 6.41 (3.020) | 7.84 (2.466)
  Nasal Blockage, Week 5, n=49, 49: number analyzed (Participants) | 49 | 49
  Nasal Blockage, Week 5, n=49, 49 | 5.66 (3.169) | 7.33 (2.489)
  Nasal Blockage, Week 9, n=48, 46: number analyzed (Participants) | 48 | 46
  Nasal Blockage, Week 9, n=48, 46 | 5.03 (3.387) | 7.22 (2.959)
  Nasal Blockage, Week 13, n=45, 39: number analyzed (Participants) | 45 | 39
  Nasal Blockage, Week 13, n=45, 39 | 4.66 (3.729) | 6.27 (3.268)
  Nasal Blockage, Week 17, n=44, 34: number analyzed (Participants) | 44 | 34
  Nasal Blockage, Week 17, n=44, 34 | 4.18 (3.556) | 5.71 (3.597)
  Nasal Blockage, Week 21, n=42, 34: number analyzed (Participants) | 42 | 34
  Nasal Blockage, Week 21, n=42, 34 | 4.04 (3.563) | 5.77 (3.397)
  Nasal Blockage, Week 25, n=42, 31: number analyzed (Participants) | 42 | 31
  Nasal Blockage, Week 25, n=42, 31 | 3.61 (3.464) | 5.81 (3.494)
  Loss of Smell, Week 1, n=49, 51 | 9.03 (1.739) | 9.22 (1.912)
  Loss of Smell, Week 2, n=49, 51 | 8.79 (1.823) | 9.02 (1.942)
  Loss of Smell, Week 5, n=49, 49: number analyzed (Participants) | 49 | 49
  Loss of Smell, Week 5, n=49, 49 | 8.28 (2.243) | 8.69 (2.511)
  Loss of Smell, Week 9, n=48, 46: number analyzed (Participants) | 48 | 46
  Loss of Smell, Week 9, n=48, 46 | 7.43 (3.192) | 8.67 (2.647)
  Loss of Smell, Week 13, n=45, 39: number analyzed (Participants) | 45 | 39
  Loss of Smell, Week 13, n=45, 39 | 7.42 (3.296) | 8.59 (2.318)
  Loss of Smell, Week 17, n=44, 34: number analyzed (Participants) | 44 | 34
  Loss of Smell, Week 17, n=44, 34 | 6.85 (3.648) | 8.18 (2.682)
  Loss of Smell, Week 21, n=42, 34: number analyzed (Participants) | 42 | 34
  Loss of Smell, Week 21, n=42, 34 | 6.74 (3.562) | 8.20 (2.835)
  Loss of Smell, Week 25, n=42, 31: number analyzed (Participants) | 42 | 31
  Loss of Smell, Week 25, n=42, 31 | 6.02 (4.069) | 7.90 (3.378)

23. Secondary Outcome: Mean Peak Nasal Inspiratory Flow (PNIF) at Weeks 2, 5, 9, 13, 17, 21, and 25
Description: Participants used a portable hand-held inspiratory flow meter to measure and record PNIF in the morning prior to taking the study medication. Three measurements were taken, and the largest measurement was recorded in the electronic diary. PNIF data is plotted and analyzed using a repeated measures model to calculate treatment difference, confidence intervals and p-values.
Time Frame: Weeks 2, 5, 9, 13, 17, 21, and 25
Population: ITT Population. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
L/min
  Week 2, n=54, 51 | 120.82 [110.59 to 131.04] | 99.66 [89.14 to 110.18]
  Week 5, n=54, 49: number analyzed (Participants) | 54 | 49
  Week 5, n=54, 49 | 127.21 [116.76 to 137.66] | 110.32 [99.39 to 121.24]
  Week 9, n=47, 46: number analyzed (Participants) | 47 | 46
  Week 9, n=47, 46 | 123.91 [110.04 to 137.77] | 116.71 [102.52 to 130.90]
  Week 13, n=45, 37: number analyzed (Participants) | 45 | 37
  Week 13, n=45, 37 | 137.50 [123.49 to 151.51] | 109.79 [94.80 to 124.78]
  Week 17, n=44, 34: number analyzed (Participants) | 44 | 34
  Week 17, n=44, 34 | 132.41 [119.40 to 145.43] | 117.02 [102.91 to 131.12]
  Week 21, n=42, 33: number analyzed (Participants) | 42 | 33
  Week 21, n=42, 33 | 143.03 [127.13 to 158.93] | 113.52 [96.28 to 130.76]
  Week 25, n=42, 32: number analyzed (Participants) | 42 | 32
  Week 25, n=42, 32 | 137.02 [121.17 to 152.87] | 110.37 [92.94 to 127.80]
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.005, repeated measures model; Mean Difference (Final Values) = 21.16, 95% CI 2-sided [6.49 to 35.83] — Week 2
Statistical Analysis 2: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.029, repeated measures model; Mean Difference (Final Values) = 16.89, 95% CI 2-sided [1.77 to 32.01] — Week 5
Statistical Analysis 3: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.472, repeated measures model; Mean Difference (Final Values) = 7.20, 95% CI 2-sided [-12.64 to 27.03] — Week 9
Statistical Analysis 4: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.009, repeated measures model; Mean Difference (Final Values) = 27.71, 95% CI 2-sided [7.19 to 48.23] — Week 13
Statistical Analysis 5: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.114, repeated measures model; Mean Difference (Final Values) = 15.40, 95% CI 2-sided [-3.80 to 34.59] — Week 17
Statistical Analysis 6: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.014, repeated measures model; Mean Difference (Final Values) = 29.51, 95% CI 2-sided [6.06 to 52.96] — Week 21
Statistical Analysis 7: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.027, repeated measures model; Mean Difference (Final Values) = 26.65, 95% CI 2-sided [3.10 to 50.21] — Week 25

24. Secondary Outcome: Olfaction Testing: Worst Nostril Score (WNS) and Mean Nostril Score (MNS) at Weeks 2, 5, 9, 13, 17, 21, and 25
Description: Sniffin'Sticks were used to assess each participant's sense of smell (olfaction). Olfaction testing results were recorded for both the right and left nostrils The worst nostril score (number of correct answers for the worst nostril) and the mean nostril score (mean number of correct answers across both nostrils) were recorded. Scores range from 0 to 12 (high score indicating normal olfactory sensation). Olfaction data are plotted and analyzed using a repeated measures model to calculate treatment difference, confidence intervals and p-values.
Time Frame: Weeks 2, 5, 9, 13, 17, 21, and 25
Population: ITT Population. Only those participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
Scores on a scale
  MNS, Week 2, n=54, 51 | 3.78 [3.29 to 4.26] | 3.68 [3.18 to 4.18]
  MNS, Week 5, n=54, 49: number analyzed (Participants) | 54 | 49
  MNS, Week 5, n=54, 49 | 4.20 [3.63 to 4.78] | 3.07 [2.46 to 3.67]
  MNS, Week 9, n=47, 45: number analyzed (Participants) | 47 | 45
  MNS, Week 9, n=47, 45 | 4.48 [3.89 to 5.07] | 3.69 [3.08 to 4.29]
  MNS, Week 13, n=45, 37: number analyzed (Participants) | 45 | 37
  MNS, Week 13, n=45, 37 | 4.39 [3.75 to 5.03] | 3.66 [2.97 to 4.35]
  MNS, Week 17, n=43, 34: number analyzed (Participants) | 43 | 34
  MNS, Week 17, n=43, 34 | 4.64 [3.93 to 5.36] | 4.26 [3.45 to 5.07]
  MNS, Week 21, n=42, 33: number analyzed (Participants) | 42 | 33
  MNS, Week 21, n=42, 33 | 4.77 [3.93 to 5.61] | 4.12 [3.19 to 5.05]
  MNS, Week 25, n=41, 32: number analyzed (Participants) | 41 | 32
  MNS, Week 25, n=41, 32 | 4.40 [3.61 to 5.18] | 3.69 [2.81 to 4.56]
  WNS, Week 2, n=54, 51 | 3.18 [2.67 to 3.69] | 2.89 [2.37 to 3.42]
  WNS, Week 5, n=54, 49: number analyzed (Participants) | 54 | 49
  WNS, Week 5, n=54, 49 | 3.72 [3.16 to 4.27] | 2.41 [1.82 to 2.99]
  WNS, Week 9, n=47, 45: number analyzed (Participants) | 47 | 45
  WNS, Week 9, n=47, 45 | 3.85 [3.21 to 4.49] | 3.17 [2.51 to 3.82]
  WNS, Week 13, n=45, 37: number analyzed (Participants) | 45 | 37
  WNS, Week 13, n=45, 37 | 3.76 [3.06 to 4.46] | 3.14 [2.38 to 3.90]
  WNS, Week 17, n=43, 34: number analyzed (Participants) | 43 | 34
  WNS, Week 17, n=43, 34 | 3.93 [3.15 to 4.70] | 3.74 [2.87 to 4.61]
  WNS, Week 21, n=42, 33: number analyzed (Participants) | 42 | 33
  WNS, Week 21, n=42, 33 | 4.16 [3.30 to 5.02] | 3.52 [2.58 to 4.47]
  WNS, Week 25, n=41, 32: number analyzed (Participants) | 41 | 32
  WNS, Week 25, n=41, 32 | 3.75 [2.93 to 4.56] | 3.30 [2.40 to 4.20]
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.790, repeated measures model; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.61 to 0.79] — MNS, Week 2
Statistical Analysis 2: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.008, repeated measures model; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [0.30 to 1.97] — MNS, Week 5
Statistical Analysis 3: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.066, repeated measures model; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.05 to 1.64] — MNS, Week 9
Statistical Analysis 4: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.127, repeated measures model; Mean Difference (Final Values) = 0.73, 95% CI 2-sided [-0.21 to 1.67] — MNS, Week 13
Statistical Analysis 5: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.481, repeated measures model; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.69 to 1.46] — MNS, Week 17
Statistical Analysis 6: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.308, repeated measures model; Mean Difference (Final Values) = 0.65, 95% CI 2-sided [-0.61 to 1.90] — MNS, Week 21
Statistical Analysis 7: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.233, repeated measures model; Mean Difference (Final Values) = 0.71, 95% CI 2-sided [-0.46 to 1.88] — MNS, Week 25
Statistical Analysis 8: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.444, repeated measures model; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.45 to 1.02] — WNS, Week 2
Statistical Analysis 9: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.002, repeated measures model; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [0.50 to 2.12] — WNS, Week 5
Statistical Analysis 10: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.143, repeated measures model; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [-0.24 to 1.60] — WNS, Week 9
Statistical Analysis 11: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.240, repeated measures model; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.42 to 1.65] — WNS, Week 13
Statistical Analysis 12: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.750, repeated measures model; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.98 to 1.35] — WNS, Week 17
Statistical Analysis 13: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.324, repeated measures model; Mean Difference (Final Values) = 0.64, 95% CI 2-sided [-0.64 to 1.91] — WNS, Week 21
Statistical Analysis 14: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.468, repeated measures model; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.77 to 1.66] — WNS, Week 25

25. Secondary Outcome: Sino-Nasal Outcome Test (SNOT)-22 Questionnaire Total Score at Week 25 (Adjusted for Week 1 Baseline)
Description: SNOT-22 questionnaire is a modification of the SNOT-20 and contains the questions (ques) related to smell and nasal obstruction. Each ques is graded with a numerical score for each response (resp); scores range from 0 for "no symptoms" to 5 for "as bad as things could be." Scores for each of the ques is summed to derive the total score for that par. at that visit. If the par. did not complete any ques at a visit, then he/she were not to have any missing values imputed, and his/her total score for that visit was set to missing. If a par. had some missing scores (but no more than 50% missing at that visit), then scores for the missing resp were imputed as the mean of the non-missing resp for that par. at that visit. The SNOT-22 total score ranges from 0 to 110, with higher scores representing a worse quality of life. Questionnaire data analysis was done using an ANCOVA to obtain the LS-means, treatment difference and confidence interval at Week 25, adjusting for Week 1 Baseline scores.
Time Frame: Week 1 (Baseline) and Week 25
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
Scores on a scale | 27.13 (2.96) | 40.36 (3.39)
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA; Mixed effects model = -13.2, 95% CI 2-sided [-22.2 to -4.22]

26. Secondary Outcome: Index Score of the EuroQoL Quality of Life-5D (EQ-5D) Questionnaire at Week 25 (Adjusting for Week 1 Baseline Scores)
Description: The EQ-5D is a standardized, 2-part questionnaire used to measure health outcomes. The first part contains descriptions of the following five components: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses to each of the five domains are measured on a 3-point scale (1-no problems, 2-some problems, and 3-severe problems). An index for the descriptive scores was derived using the general European weights, obtained for each of the countries in this study. Index scores were derived for each participant at each time point by taking sum of weights. Index score ranges from -0.718 to 1, with lower scores indicating poor health. ANCOVA model with treatment, Baseline (Week 1 scores) and country as factors was used to calculate treatment difference and confidence intervals at Week 25.
Time Frame: Week 1 (Baseline) and Week 25
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
Scores on a scale | 0.91 (0.02) | 0.91 (0.02)
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.06 to 0.07]

27. Secondary Outcome: VAS Score of the EQ-5D Questionnaire at Week 25 (Adjusting for Week 1 Baseline Scores)
Description: The EQ-5D is a standardized, 2-part questionnaire used to measure health outcomes. The second part of the questionnaire is a VAS question, requiring the participant to self rate his/her health score on a scale of 0 (worst imaginable health state) to 100 (best imaginable health state). ANCOVA model with treatment, Baseline (Week 1 scores) and country as factors was used to calculate treatment difference and confidence intervals at Week 25.
Time Frame: Week 1 (Baseline) and Week 25
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 54 | 51
Scores on a scale | 81.13 (2.30) | 75.45 (2.64)
Statistical Analysis 1: Comparison: Mepolizumab 750 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 5.68, 95% CI 2-sided [-1.33 to 12.68]

28. Secondary Outcome: Systemic Clearance of Mepolizumab 750 mg
Description: Blood samples were collected for the assessment of systemic clearance at Weeks 1, 2, 5, 9, 13, and 25. Systemic Clearance (CL) is estimated using a population-Pharmacokinetic model incorporating all available data points from all participants. Individual values were estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, and 25
Population: Pharmacokinetic (PK) Population: participants in the Safety Population for whom at least one PK sample was obtained and analyzed.
Measure: Mean (Standard Deviation); unit: Liters per day
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 52
Liters per day | 0.250 (0.0659)

29. Secondary Outcome: Volume of Distribution of Mepolizumab 750 mg
Description: Volume of distribution at steady-state was derived from pharmacokinetic parameter estimates of a population pharmacokinetic model. Blood samples were collected for analysis of volume of distribution at Weeks 1, 2, 5, 9, 13, and 25. All available concentrations at all available datapoints from all participants were incorporated into the model. Individual values were estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 52
Liters | 8.387 (2.0062)

30. Secondary Outcome: Bodyweight-adjusted Clearance
Description: Clearance is the volume of plasma that would contain the amount of drug excreted per day. Blood samples were collected for the assessment of bodyweight-adjusted clearance at Weeks 1, 2, 5, 9, 13, and 25. Clearance was estimated using a population-pharmacokinetic model incorporating all available data points from all participants. Individual values were estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per day
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 52
Liters per day | 0.2170 (0.009547)

31. Secondary Outcome: Steady-State Volume of Distribution
Description: Steady-state volume of distribution is the blood and tissue volume into which a drug is distributed and the relative binding of drug to protein in these spaces. Blood samples were collected for the assessment of steady-state volume of distribution at Weeks 1, 2, 5, 9, 13, and 25. Steady-state volume of distribution was estimated using a population-pharmacokinetic model incorporating all available data points from all participants. Individual values were estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 52
Liters | 7.0958 (0.3226)

32. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax), Average Concentration (Cav[0-inf]), and Steady State Maximum Observed Plasma Drug Concentration (Cmax SS)
Description: Blood samples were collected for the assessment of Cmax, Cav(0-inf), and Cmax SS at Weeks 1, 2, 5, 9, 13, and 25. These parameters were estimated using a population-pharmacokinetic model incorporating all available data points from all participants. Individual values were estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Micrograms per milliliter
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 52
Micrograms per milliliter
  Cmax | 193.22 (7.8536)
  Cav(0-inf) | 123.45 (5.4324)
  Cmax SS | 268.40 (10.3703)

33. Secondary Outcome: Area Under the Plasma Drug Concentration Versus Time Curve From Time 0 Extrapolated to Infinite Time (AUC[0-inf])
Description: Blood samples were scheduled to be collected for the assessment of AUC(0-inf) at Weeks 1, 2, 5, 9, 13, and 25 AUC[0-inf] is derived from individual systemic clearance estimates using the expression AUC[0-inf] = Dose/CL. Hence all data are incorporated into the estimation of CL and by implication AUC[0-inf].
Time Frame: Weeks 1, 2, 5, 9, 13, and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Day*Microgram per milliliter
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 52
Day*Microgram per milliliter | 3456.69 (152.11)

34. Secondary Outcome: Half-life (Alpha) and Half-life (Beta)
Description: Half-life (Alpha) is the rate of decline in plasma concentrations due to the process of drug redistribution from the central to the peripheral compartment and half-life (Beta ) is the rate of decline due to the process of drug elimination due to metabolism. Blood samples were collected for the assessment of half-life (Alpha) and half-life (Beta) at Weeks 1, 2, 5, 9, 13, and 25. Half-life was estimated using a population-pharmacokinetic model incorporating all available data points from all participants. Individual values were estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 52
Days
  Half-life (Alpha) | 1.5456 (0.4108)
  Half-life (Beta) | 24.1258 (1.0250)

35. Secondary Outcome: Pharmacokinetic/Pharmacodynamic (PK/PD) Model Derived Baseline
Description: Blood samples were collected for the assessment of PK/PD model derived Baseline at Weeks 1, 2, 5, 9, 13, 17, 21 and 25. An exploratory Emax direct response model was fitted to serial blood eosinophil count data (including placebo) using model-predicted mepolizumab concentrations (with zero imputed for placebo treated participants). All available blood eosinophil count data were incorporated into the model. Individual values were estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21 and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Giga units per liter
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 104
Giga units per liter | 0.4231 (0.02873)

36. Secondary Outcome: PK/PD Model Derived Coefficient of Variation of Baseline (CV[Baseline]), Variation of Maximal Effect of Drug (CV[Emax]), and Residual
Description: A residual is the difference between the observed and predicted values. Blood samples were collected for the assessment of PK/PD model derived CV(Baseline), CV(Emax), and residual at Weeks 1, 2, 5, 9, 13, 17, 21 and 25. An exploratory Emax direct response model was fitted to serial blood eosinophil count data (including placebo) using model-predicted mepolizumab concentrations (with zero imputed for placebo treated subjects). All available datapoints were incorporated into the model. Individual values are estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21 and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of variation
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 104
Percentage of variation
  CV(Baseline) | 51.9951 (6.5318)
  CV(Emax) | 52.8910 (6.6193)
  Residual | 41.3787 (1.3763)

37. Secondary Outcome: PK/PD Model Derived Half Maximal Effective Drug Concentration (EC50)
Description: Blood samples were collected for the assessment of PK/PD model derived EC50 at Weeks 1, 2, 5, 9, 13, 17, 21 and 25. An exploratory Emax direct response model was fitted to serial blood eosinophil count data (including placebo) using model-predicted mepolizumab concentrations (with zero imputed for placebo treated participants). All available datapoints were incorporated into the model. Individual values are estimated from the model as post-hoc values after incorporating between-partcipant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21 and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Microgram per liter
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 104
Microgram per liter | 4.4303 (0.4404)

38. Secondary Outcome: PK/PD Model Derived Maximum Inhibition
Description: Blood samples were collected for the assessment of Maximum Inhibition at Weeks 1, 2, 5, 9, 13, 17, 21 and 25. An exploratory Emax direct response model was fitted to serial blood eosinophil count data (including placebo) using model-predicted mepolizumab concentrations (with zero imputed for placebo treated participants). All available datapoints were incorporated into the model. Individual values are estimated from the model as post-hoc values after incorporating between-participant variability.
Time Frame: Weeks 1, 2, 5, 9, 13, 17, 21 and 25
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of inhibition
Arm/Group | Mepolizumab 750 mg
Number analyzed (Participants) | 104
Percentage of inhibition | 90.0748 (1.0096)

39. Secondary Outcome: Number of Participants With Positive Immunogenicity (Anti-mepolizumab Antibody Testing)
Description: Blood samples were collected at Week 1 pre-dose, Week 5 pre-dose, Week 13 pre-dose and Week 25 (4 weeks post last dose) for anti-mepolizumab antibody testing using a validated electrochemiluminescent (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'.
Time Frame: Week 1 pre-dose, Week 5 pre-dose, Week 13 pre-dose and Week 25 (4 weeks post last dose)
Population: Safety Population. One participant randomized to mepolizumab took placebo in error. Thus, "N" for the placebo arm of the SP is greater than for the ITT Population. Participants available at the specified time points (represented by n=X, X) were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 750 mg | Placebo
Number analyzed (Participants) | 53 | 52
Participants
  Week 1, pre-dose, n=53, 52 | 0 | 2
  Week 5, pre-dose, n=53, 50: number analyzed (Participants) | 53 | 50
  Week 5, pre-dose, n=53, 50 | 0 | 2
  Week 13, pre-dose, n=45, 40: number analyzed (Participants) | 45 | 40
  Week 13, pre-dose, n=45, 40 | 0 | 2
  Week 25, 4 weeks post last dose, n=40, 31: number analyzed (Participants) | 40 | 31
  Week 25, 4 weeks post last dose, n=40, 31 | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the first dose of flixonase administration (at the start of the Run-in Period) up to the end of the study (up to 11 months)
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all enrolled participants who received at least one dose of study medication.One participant randomized to mepolizumab took placebo in error. Thus, "N" for the placebo arm of the SP is greater than for the ITT Population.
Arm/Group | Mepolizumab 750 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 32/53 | 38/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 750 mg (N=53) | Placebo (N=52)
Ear pain (Ear and labyrinth disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 2 | 4
Fatigue (General disorders) | 1 | 5
Influenza (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 10 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Headache (Nervous system disorders) | 13 | 20
Sinus headache (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Pyrexia (General disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
Part B was removed due to the low numbers of participants enrolling into Part B. GSK determined it was no longer feasible to achieve a meaningful number of participants and therefore recruitment into this portion of the study was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.